CLINICAL TRIAL: NCT03488719
Title: A Phase 1 Study to Examine Pharmacodynamic Interaction Between Tesofensine and Metoprolol on 24-hours Mean Heart Rate
Brief Title: A Study to Examine the Effect of Tesofensine and Metoprolol on the 24-hour Mean Heart Rate
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Saniona (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: TM004
Record Dates: First submitted 2018-03-12; First posted 2018-04-05 (Actual); Results first posted 2024-02-09 (Actual); Last update posted 2024-02-09 (Actual); Status verified 2023-06

CONDITIONS: Phase 1
MeSH Terms: interventions — Metoprolol

STUDY DESIGN:
Intervention Model Description: Each subject will participate in a Screening Period (Day 28 to Day 3), a Baseline Period (Day -2 to Day -1) and a Treatment Period (Day 1 to Day 24) and will have two Follow-up phone calls (Day 30 and Day 50).
Who Masked: Participant, Care Provider, Investigator
Masking Description: Tesofensine dosing will be performed open-label. Metoprolol dosing will be performed "single-blind".
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Cohort 1 (Tesofensine 0.25mg) (Experimental): Tesofensine 0.25 mg once daily for 23 days (loading dose of 1.0 mg for the first 3 days), plus a single dose of 25 mg, 50 mg or 100 mg metoprolol extended release (ER) in random order on Day 15, Day 18 and Day 21, respectively.
  Interventions: Drug: Metoprolol Succinate 25 MG; Drug: Metoprolol Succinate 50 MG; Drug: Metoprolol Succinate 100 MG
- Cohort 2 (Tesofensine 0.50mg) (Experimental): Tesofensine 0.50 mg once daily for 23 days (loading dose of 2.0 mg for the first 3 days), plus a single dose of 25 mg, 50 mg or 100 mg metoprolol extended release (ER) in random order on Day 15, Day 18 and Day 21, respectively.
  Interventions: Drug: Metoprolol Succinate 25 MG; Drug: Metoprolol Succinate 50 MG; Drug: Metoprolol Succinate 100 MG
- Cohort 3 (Tesofensine 0.75mg) (Experimental): Tesofensine 0.75 mg (0.25 mg + 0.50 mg) once daily for 23 days (loading dose of 2.0 mg [4 tablets of 0.50 mg] for the first 5 days), plus a single dose of 25 mg, 50 mg or 100 mg metoprolol extended release (ER) in random order on Day 15, Day 18 and Day 21, respectively.
  Interventions: Drug: Metoprolol Succinate 25 MG; Drug: Metoprolol Succinate 50 MG; Drug: Metoprolol Succinate 100 MG

INTERVENTIONS:
Drug: Metoprolol Succinate 25 MG — A single dose of 25 mg metoprolol ER in the morning of Day 15, Day 18 or Day 21 approximately 30 minutes after start of a standard breakfast and together with the tesofensine dose.
Drug: Metoprolol Succinate 50 MG — A single dose of 50 mg metoprolol ER in the morning of Day 15, Day 18 or Day 21 approximately 30 minutes after start of a standard breakfast and together with the tesofensine dose.
Drug: Metoprolol Succinate 100 MG — A single dose of 100 mg metoprolol ER in the morning of Day 15, Day 18 or Day 21, approximately 30 minutes after start of a standard breakfast and together with the tesofensine dose.

SUMMARY:
A Phase 1 Study to Examine Pharmacodynamic Interaction Between Tesofensine and Metoprolol on 24-hours Mean Heart Rate

DETAILED DESCRIPTION:
In this study, the dose-response relationship between tesofensine and metoprolol will be examined and thus the optimal dose of metoprolol to mitigate the effects of tesofensine on heart rate (HR) will be determined. HR is the primary endpoint because in the previous studies it has been shown to be the most affected safety endpoint by the effects of tesofensine.

After enrolment of 37 subjects, 2 Subjects (0115 and 0147) in dose cohort 2 experienced prolonged tachycardia (> 120 beats per minute (bpm) lasting for 30 min) documented in Holter Electrocardiogram (ECG) recording (a stopping criteria of the study). Therefore, the study was temporarily halted on 22 November 2018. Subsequent to the temporary halt, Saniona reviewed all the available data in January and February 2019 and determined that the results obtained from the completed participants were sufficiently robust to answer the questions for which the trial was designed. Therefore, Saniona decided to permanently end the trial on 20 February 2019.

ELIGIBILITY:
Inclusion Criteria:

1. Subject voluntarily agreed to participate in this study and signed an Independent Ethics Committee (IEC)-approved informed consent prior to performing any of the Screening procedures.
2. Male and female subjects between 18 to 60 years of age, inclusive, at Screening.
3. Overweight and obese subjects with a body mass index (BMI) between ≥ 27 and < 40 kg/m2 at Screening but otherwise healthy.
4. Non-smokers (or other nicotine use) as determined by history (no nicotine use over the past 6 months) and by urine cotinine concentration (< 500 ng/mL) at Screening and admission.
5. No clinically relevant deviation or finding in pre-study medical evaluation (medical history, physical examination, vital signs, 12-lead electrocardiogram (ECG) and clinical laboratory evaluations).
6. Hemoglobin A1c (HbA1c) < 6.5% at Screening.
7. Subject was willing to adhere to the contraception requirements details.

Exclusion Criteria:

1. Subject had history or evidence of any clinically significant cardiovascular, gastrointestinal, endocrinologic, hematologic, hepatic, immunologic, metabolic (e.g., diabetes, metabolic acidosis), urologic, pulmonary (e.g., asthma or chronic obstructive pulmonary disease), neurologic, dermatologic, psychiatric, renal, and/or other major disease or malignancy as judged by the Investigator.
2. Subject had any disorder that would interfere with the absorption, distribution, metabolism or excretion of drugs.
3. Subject had a clinically significant abnormality following the Investigator's review of the physical examination, ECG and clinical study protocol (CSP)-defined clinical laboratory tests at Screening or admission to the clinical unit or had any concurrent disease or condition that, in the opinion of the Investigator, would make the subject unsuitable for participation in the clinical study. One re-test was allowed, if (a) test result(s) was outside the limits.
4. History or presence of liver disease or liver injury, as indicated by abnormal liver function tests including:

   * Aspartate aminotransferase (AST) > 1.2 x upper limit of normal (ULN)
   * Alanine aminotransferase (ALT) > 1.1 x upper limit of normal (ULN)
5. Subject had a pulse < 50 or > 90 beats per minute (bpm); systolic blood pressure (SBP) < 90 mmHg or > 140 mmHg; diastolic blood pressure (DBP) < 50 mmHg or > 90 mmHg (using the mean of triplicate measurements) at Screening or admission. One re-test was allowed, if (a) test result(s) was outside these limits.
6. History of any clinically significant cardiac arrhythmia. Subject had a corrected QT interval using Fridericia's formula (QTcF) interval > 450 msec or 2nd or 3rd degree atrioventricular (AV) block, high-grade sinoatrial block or PQ interval > 0.24 seconds at Screening (using the mean of triplicate measurements). If a mean ECG parameter of a triplicate ECG exceeded the limits above, an additional triplicate ECG could have been taken. If this also gave an abnormal result, the subject was excluded. Also, the following cardiac conditions led to exclusion of the subjects: Untreated heart failure (pulmonary oedema, impaired blood flow or hypotension) and continuous or intermittent treatment leading to an increased contractility of the heart muscle (beta-receptor agonism); sick sinus syndrome; cardiogenic shock; severe peripheral arterial circulatory disturbances.
7. Had a creatinine value exceeding the ULN.
8. Subject had a positive test for hepatitis B surface antigen (HBsAg), or hepatitis B core antibody (indicative of active hepatitis B), hepatitis A virus antibodies (immunoglobulin M), hepatitis C virus (HCV) antibodies or human immunodeficiency virus (HIV) type 1 and/or type 2 antibodies.
9. Use of any prescribed or non-prescribed drugs (including vitamins, natural and herbal remedies, e.g., St. John's Wort) in the 2 weeks prior to admission or 5 half-lives of the drug, whichever was longer, except for the occasional use of paracetamol (up to 2 g/day) or other non-steroidal anti-inflammatory drugs (NSAIDs) and hormonal contraception for female subjects.
10. Subject had history of alcohol and/or illicit drug abuse within 2 years of entry.
11. Subject had positive urine drug test (e.g., cocaine, amphetamines, barbiturates, opiates, benzodiazepines, cannabinoids) or alcohol test at Screening or at admission.
12. History of drinking > 168 g (males) and > 84 g (females) pure alcohol per week (10 g pure alcohol = 259 mL of beer [5%] or 35 mL of spirits [35%] or 100 mL of wine [12%] within 3 months prior to admission to the clinical unit.
13. Subject consumed more than 600 mg caffeine per day (e.g., more than 3 cups of coffee containing 200 mg caffeine per cup) within the 4 weeks before admission or the subject was unwilling to avoid consumption of coffee and caffeine-containing beverages within 48 hours prior to admission until discharge from the clinical unit.
14. Subject was unwilling to avoid use of alcohol or alcohol-containing foods, medications or beverages, within 48 hours prior to Screening and from admission until discharge from the clinical unit.
15. Any significant blood loss, donated 1 unit (450 mL) of blood or more, or received a transfusion of any blood or blood products within 60 days, or donated plasma within 7 days prior to the admission to the clinical unit.
16. Participation in any clinical study within 3 months or 5 half-lives of the drug, whichever was longer, prior to the expected date of IMP administration, or participation in more than 3 clinical studies within 12 months.
17. Subject with a relevant history or with a present psychiatric disorder, including depression, suicidal ideation, or eating disorders (e.g., bulimia or anorexia nervosa). Subjects with a medical history of relevant psychiatric disorders or known and relevant family history or evidence of anxiety disorders or depression as judged by the Investigator using the Generalized Anxiety Disorder Assessment-7 (GAD-7) and Patient Health Questionnaire-9 (PHQ-9) at Screening. Any of the following led to exclusion of the subject:

    * Subject had a GAD-7 mood scale score ≥ 10.
    * Subject had a score ≥ 10 on the PHQ-9 questionnaire.
    * Subject selected a response of "1, 2 or 3" to question number 9 on the PHQ-9 questionnaire regarding potential for suicidal thoughts or ideation (independent of the total score of the PHQ-9).
18. Use of any agent used for weight loss within the last 3 months.
19. More than 5% weight loss within the last 3 months.
20. Hypo- or hyperthyroidism.
21. Subject was pregnant or lactating.
22. Subject was unwilling to abstain from vigorous exercise from 48 hours prior to admission until discharge.
23. Subject had a history of hypersensitivity to the Investigational medicinal products (IMPs) or any of the excipients or to medicinal products with similar chemical structures.
24. Any contraindication for metoprolol, e.g., severe peripheral arterial disease, untreated pheochromocytoma, concomitant intravenous administration of calcium antagonists of verapamil and diltiazem, due to the risk of hypotension, atrioventricular (AV) conduction disturbances, or left ventricular insufficiency.
25. Subject had lactose intolerance or a rare hereditary problem of fructose intolerance, glucose galactose malabsorption or sucrase isomaltase insufficiency.
26. Subject was unable to understand and communicate in German language or to understand the protocol requirements, instructions and study-related restrictions, the nature, scope and possible consequences of the clinical study or was unlikely to comply with the study requirements; e.g., uncooperative attitude and improbability of completing the clinical study.
27. Subject had previously been enrolled in this clinical study.
28. Vulnerable subjects defined as individuals whose willingness to volunteer in a clinical study may be unduly influenced by the expectation, whether justified or not, of benefits associated with participation, or of a retaliatory response from senior members of a hierarchy in case of refusal to participate (e.g., persons in detention, minors and those incapable of giving consent).
29. Subject was the Investigator or any Sub-Investigator, research assistant, pharmacist, study coordinator, other staff or relative thereof directly involved in the conduct of the study or employee of the Sponsor or Parexel.
30. Poor or ultra-rapid cytochrome P450 2D6 (CYP2D6) metabolizer.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 37 (Actual)
Dates: Start 2018-07-11 (Actual); Primary Completion 2019-06-06 (Actual); Study Completion 2019-06-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kim Krogsgaard, MD, DMSc, Study Director — Saniona
Locations (1):
- Parexel International GmbH; Early Phase Clinical Unit Berlin, Berlin, Germany

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Cohort 1 (Tesofensine 0.25mg) | Cohort 2 (Tesofensine 0.50mg) | Cohort 3 (Tesofensine 0.75mg)
Started | 9 | 16 | 12
Metoprolol 25 mg | 9 | 13 | 5
Metoprolol 50 mg | 9 | 13 | 6
Metoprolol 100 mg | 9 | 13 | 5
Completed | 9 | 12 | 5
Not Completed | 0 | 4 | 7
Not completed — Adverse Event | 0 | 4 | 2
Not completed — Other | 0 | 0 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1 (Tesofensine 0.25mg) | Cohort 2 (Tesofensine 0.50mg) | Cohort 3 (Tesofensine 0.75mg) | Total
Number analyzed (Participants) | 9 | 16 | 12 | 37
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.4 (10.68) | 43.1 (11.61) | 43.8 (9.74) | 43.9 (10.55)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 8 | 5 | 17
  Male | 5 | 8 | 7 | 20
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 9 | 16 | 12 | 37
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 9 | 16 | 12 | 37
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Height [Mean (Standard Deviation); unit: cm] | 174.1 (10.91) | 171.1 (9.84) | 170.1 (6.49) | 171.5 (9.06)
Weight [Mean (Standard Deviation); unit: kg] | 95.52 (11.602) | 88.56 (9.801) | 91.08 (10.925) | 91.07 (10.685)

OUTCOME MEASURES:

1. Primary Outcome: Dose of Metoprolol Resulting in no Change in Mean Heart Rate Over 24 Hours (M24HR)
Description: The dose of metoprolol which resulted in no change relative to baseline in mean heart rate over 24 hours (M24HR) for each respective dose of tesofensine was calculated from a dose response relationship with the log-dose of metoprolol as independent variable and change in M24HR induced by various doses of metoprolol given to subjects on steady-state dose of tesofensine as the dependent variable. The dose for no change in M24HR derived from above calculation and the corresponding 95% confidence interval (CI) is presented for each dose of tesofensine. The result in this endpoint is not an arithmetic mean, but the model derived estimated dose from the model. Mitigating dose was estimated using a linear regression modelling mean change from pre-tesofensine baseline (Day -1) of M24HR as a function of the log metoprolol dose.
Time Frame: Day -1 to Day 23
Population: Pharmacodynamic (PD) Population: All randomized subjects with at least HR assessments (24 Hour Holter) on Baseline (Day -2 to -1) and on at least 2 Visits out of, Day 15, Day 18 and Day 21 without any major protocol deviations which could have influenced the PD parameters.
Measure: Mean (95% Confidence Interval); unit: mg
Arm/Group | Cohort 1 (Tesofensine 0.25mg) | Cohort 2 (Tesofensine 0.50mg) | Cohort 3 (Tesofensine 0.75mg)
Number analyzed (Participants) | 9 | 13 | 6
mg | 10.04 [0.01 to 34.26] | 60.95 [35.27 to 99.43] | 147.91 [61.28 to 362.29]

2. Secondary Outcome: Mean Heart Rate Over 24 Hours (M24HR) at Baseline (Day -1) and Days 14, 17, 20 and 23
Description: M24HR at Baseline (Day -1) and Days 14, 17, 20 and 23.
Time Frame: Baseline (Day -1), Days 14, 17, 20 and 23
Population: Pharmacodynamic population required heart rate (HR) at baseline and at least 2 visits out of Day 15, Day 18, Day 21, thus subjects discontinued before Day 18 were excluded. The number of participants listed below is the number of subjects with an assessment at the specified time point.
Measure: Mean (Standard Deviation); unit: bpm
Arm/Group | Cohort 1 (Tesofensine 0.25mg) | Cohort 2 (Tesofensine 0.50mg) | Cohort 3 (Tesofensine 0.75mg)
Number analyzed (Participants) | 9 | 13 | 6
bpm
  Baseline | 73.4 (8.47) | 73.1 (5.48) | 74.3 (5.82)
  Day 14 | 72.6 (8.17) | 76.5 (6.98) | 81.3 (4.97)
  Day 17 | 75.1 (10.93) | 78.2 (5.85) | 84.7 (8.31)
  Day 20: number analyzed (Participants) | 9 | 13 | 5
  Day 20 | 75.7 (9.33) | 80.9 (5.84) | 83.2 (7.98)
  Day 23: number analyzed (Participants) | 9 | 12 | 5
  Day 23 | 78.8 (10.41) | 84.3 (8.59) | 85.4 (7.16)

3. Secondary Outcome: Mean Heart Rate Over 24 Hours (M24HR) on Days 15, 18 or 21
Description: M24HR following each of the 3 metoprolol doses (M24HR on Days 15, 18 or 21).
Time Frame: Days 15, 18, or 21
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: bpm
Arm/Group | Cohort 1 (Tesofensine 0.25mg) | Cohort 2 (Tesofensine 0.50mg) | Cohort 3 (Tesofensine 0.75mg)
Number analyzed (Participants) | 9 | 13 | 6
bpm
  Metoprolol 25 mg | 71.1 (9.45) | 76.5 (7.68) | 80.0 (7.71)
  Metoprolol 50 mg | 69.6 (9.40) | 73.9 (5.75) | 80.8 (7.83)
  Metoprolol 100 mg: number analyzed (Participants) | 9 | 12 | 5
  Metoprolol 100 mg | 69.2 (9.46) | 70.7 (6.05) | 73.6 (3.91)

4. Secondary Outcome: Change in Mean Heart Rate Over 24 Hours (M24HR) Between Pre-tesofensine Baseline (Day -1) and After Tesofensine Alone (Day 14, Day 17, Day 20 and Day 23)
Description: Change in M24HR between pre-tesofensine baseline (Day -1) and after tesofensine alone (Day 14, Day 17, Day 20 and Day 23)
Time Frame: Baseline (Day -1), Day 14, Day 17, Day 20, Day 23
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: bpm
Arm/Group | Cohort 1 (Tesofensine 0.25mg) | Cohort 2 (Tesofensine 0.50mg) | Cohort 3 (Tesofensine 0.75mg)
Number analyzed (Participants) | 9 | 13 | 6
bpm
  Change at Day 14 | -0.9 (2.20) | 3.5 (4.50) | 7.0 (5.69)
  Change at Day 17 | 1.7 (5.32) | 5.2 (4.56) | 10.3 (6.44)
  Change at Day 20: number analyzed (Participants) | 9 | 13 | 5
  Change at Day 20 | 2.2 (3.31) | 7.8 (3.21) | 10.0 (6.48)
  Change at Day 23: number analyzed (Participants) | 9 | 12 | 5
  Change at Day 23 | 5.3 (5.34) | 11.8 (6.62) | 12.2 (6.83)

5. Secondary Outcome: Change in Mean Heart Rate Over 24 Hours (M24HR) Values After Tesofensine Co-administered With Metoprolol
Description: Change in M24HR values after tesofensine co-administered with metoprolol. As the three metoprolol doses were given in a random order these results are not reported as Day 15, Day 18 and Day 21 but instead as change from matched day.
Time Frame: Day 15, Day 18, Day 21
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: bpm
Arm/Group | Cohort 1 (Tesofensine 0.25mg) | Cohort 2 (Tesofensine 0.50mg) | Cohort 3 (Tesofensine 0.75mg)
Number analyzed (Participants) | 9 | 13 | 6
bpm
  Metoprolol 25 mg: number analyzed (Participants) | 9 | 13 | 5
  Metoprolol 25 mg | 2.7 (2.87) | -2.9 (2.25) | -2.2 (2.05)
  Metoprolol 50 mg | -4.8 (2.77) | -4.8 (2.89) | -4.7 (2.42)
  Metoprolol 100 mg: number analyzed (Participants) | 9 | 13 | 5
  Metoprolol 100 mg | -6.0 (3.50) | -6.9 (2.50) | -7.6 (2.30)

6. Secondary Outcome: Maximum and Minimum Heart Rate of 24 Hours (HRmax and HRmin) Values After Tesofensine Alone (Day 14, Day 17, Day 20 and Day 23)
Description: Maximum and minimum heart rate of 24 hours (HRmax and HRmin) values after tesofensine alone (Day 14, Day 17, Day 20 and Day 23)
Time Frame: Day 14, Day 17, Day 20 and Day 23
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: bpm
Arm/Group | Cohort 1 (Tesofensine 0.25mg) | Cohort 2 (Tesofensine 0.50mg) | Cohort 3 (Tesofensine 0.75mg)
Number analyzed (Participants) | 9 | 13 | 6
bpm
  HRmax Day 14 | 114.4 (11.53) | 117.5 (10.43) | 124.2 (17.79)
  HRmax Day 17 | 119.2 (19.47) | 124.6 (11.57) | 126.2 (17.63)
  HRmax Day 20;: number analyzed (Participants) | 9 | 13 | 5
  HRmax Day 20; | 117.0 (18.83) | 125.2 (12.21) | 131.0 (20.36)
  HRmax Day 23: number analyzed (Participants) | 9 | 12 | 5
  HRmax Day 23 | 125.6 (10.19) | 134.5 (12.77) | 133.6 (17.97)
  HRmin Day 14 | 54.2 (6.51) | 56.7 (5.78) | 59.5 (4.42)
  HRmin Day 17 | 54.1 (7.11) | 58.5 (4.86) | 60.2 (6.74)
  HRmin Day 20: number analyzed (Participants) | 9 | 13 | 5
  HRmin Day 20 | 55.0 (6.36) | 58.9 (5.53) | 60.6 (6.95)
  HRmin Day 23: number analyzed (Participants) | 9 | 12 | 5
  HRmin Day 23 | 56.8 (7.60) | 59.7 (5.69) | 61.6 (6.11)

7. Secondary Outcome: Maximum Heart Rate (HRmax) and Minimum Heart Rate (HRmin) Values After Tesofensine Co-administered With Metoprolol (Day 15, Day 18 and Day 21)
Time Frame: Day 15, Day 18, Day 21
Population: Pharmacodynamic population required heart rate (HR) at baseline and at least 2 visits out of Day 15, Day 18, Day 21, thus subjects discontinued before Day 18 were excluded. The number of participants listed below is the number of subjects with an assessment at given time point.
Measure: Mean (Standard Deviation); unit: bpm
Arm/Group | Cohort 1 (Tesofensine 0.25mg) | Cohort 2 (Tesofensine 0.50mg) | Cohort 3 (Tesofensine 0.75mg)
Number analyzed (Participants) | 9 | 13 | 6
bpm
  Metoprolol 25 mg; HR max: number analyzed (Participants) | 9 | 13 | 5
  Metoprolol 25 mg; HR max | 107.3 (11.93) | 117.8 (14.32) | 120.0 (11.73)
  Metoprolol 25 mg; HR min: number analyzed (Participants) | 9 | 13 | 5
  Metoprolol 25 mg; HR min | 53.7 (8.06) | 56.7 (5.89) | 57.4 (3.51)
  Metoprolol 50 mg; HR max | 113.2 (19.90) | 118.5 (10.24) | 125.0 (14.14)
  Metoprolol 50 mg; HR min | 51.9 (6.09) | 55.9 (4.65) | 55.7 (5.43)
  Metoprolol 100 mg; HR max: number analyzed (Participants) | 9 | 13 | 5
  Metoprolol 100 mg; HR max | 112.7 (19.89) | 111.9 (9.42) | 114.0 (12.27)
  Metoprolol 100 mg; HR min: number analyzed (Participants) | 9 | 13 | 5
  Metoprolol 100 mg; HR min | 51.7 (7.68) | 52.9 (4.66) | 55.6 (4.56)

8. Secondary Outcome: Mean Heart Rate (HR) During a Designated Quiet Hour and a Designated Period After Tesofensine Alone (Day 14, Day 17, Day 20 and Day 23)
Time Frame: From 12 to 13 hours post-dose on Day 14, Day 17, Day 20 and Day 23
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: bpm
Arm/Group | Cohort 1 (Tesofensine 0.25mg) | Cohort 2 (Tesofensine 0.50mg) | Cohort 3 (Tesofensine 0.75mg)
Number analyzed (Participants) | 9 | 13 | 6
bpm
  Day 14 | 70.0 (9.99) | 71.4 (9.52) | 77.8 (10.50)
  Day 17 | 73.4 (12.57) | 72.9 (7.45) | 80.3 (11.48)
  Day 20: number analyzed (Participants) | 9 | 13 | 5
  Day 20 | 73.0 (11.15) | 75.8 (8.33) | 77.8 (8.38)
  Day 23: number analyzed (Participants) | 9 | 12 | 5
  Day 23 | 75.7 (12.24) | 76.8 (10.63) | 77.8 (7.40)

9. Secondary Outcome: Mean Heart Rate (HR) During a Designated Quiet Hour and a Designated Period After Tesofensine Co-administered With Metoprolol (Day 15, Day 18 and Day 21)
Time Frame: From 12 to 13 hours post-dose on Day 15, Day 18, or Day 21
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: bpm
Arm/Group | Cohort 1 (Tesofensine 0.25mg) | Cohort 2 (Tesofensine 0.50mg) | Cohort 3 (Tesofensine 0.75mg)
Number analyzed (Participants) | 9 | 13 | 6
bpm
  Metoprolol 25 mg: number analyzed (Participants) | 9 | 13 | 5
  Metoprolol 25 mg | 66.8 (11.45) | 70.5 (8.75) | 77.6 (9.21)
  Metoprolol 50 mg | 65.7 (10.20) | 68.8 (7.91) | 74.2 (10.19)
  Metoprolol 100 mg: number analyzed (Participants) | 9 | 13 | 5
  Metoprolol 100 mg | 65.4 (10.99) | 65.6 (8.14) | 68.4 (7.33)

10. Secondary Outcome: Heart Rate (HR) After at Least 10 Minutes Rest Before Each Pharmacokinetic (PK) Sampling Time Point or the Corresponding Time Point (Day -1, Day 13 [Pre-dose Only], Day 14, Day 15, Day 17, Day 18, Day 20, Day 21 and Day 23)
Time Frame: Day -1, Day 13 [pre-dose only], Day 14, Day 15, Day 17, Day 18, Day 20, Day 21 and Day 23
Population: All subjects included in the study and dosed with investigational medicinal product (IMP) were included in the safety population. The number of participants listed below is the number of subjects with an assessment at the specified time point.
Measure: Mean (Standard Deviation); unit: bpm
Arm/Group | Cohort 1 (Tesofensine 0.25mg) | Cohort 2 (Tesofensine 0.50mg) | Cohort 3 (Tesofensine 0.75mg)
Number analyzed (Participants) | 9 | 16 | 12
bpm
  Day -1/predose | 62.11 (6.579) | 63.14 (7.703) | 65.71 (7.051)
  Day -1/2h postdose | 70.03 (7.317) | 71.65 (8.236) | 70.18 (9.287)
  Day -1/4h postdose | 65.60 (8.408) | 65.71 (8.705) | 66.87 (8.109)
  Day -1/8h postdose | 64.26 (7.590) | 65.38 (7.077) | 65.93 (7.195)
  Day -1/12h postdose | 72.13 (10.416) | 68.17 (6.511) | 71.08 (9.917)
  Day 13/predose: number analyzed (Participants) | 9 | 14 | 7
  Day 13/predose | 64.89 (6.680) | 71.48 (8.783) | 74.11 (7.645)
  Day 14/predose: number analyzed (Participants) | 9 | 14 | 7
  Day 14/predose | 62.41 (6.929) | 63.98 (6.973) | 70.01 (7.574)
  Day 14/2h postdose: number analyzed (Participants) | 9 | 14 | 7
  Day 14/2h postdose | 66.00 (9.106) | 70.11 (8.787) | 72.53 (8.269)
  Day 14/4h postdose: number analyzed (Participants) | 9 | 14 | 7
  Day 14/4h postdose | 62.81 (7.803) | 69.03 (9.568) | 72.03 (9.966)
  Day 14/8h postdose: number analyzed (Participants) | 9 | 14 | 7
  Day 14/8h postdose | 64.57 (8.509) | 69.76 (9.156) | 73.49 (7.267)
  Day 14/12h postdose: number analyzed (Participants) | 9 | 14 | 7
  Day 14/12h postdose | 70.19 (10.114) | 72.65 (9.286) | 80.17 (9.304)
  Day 17/predose: number analyzed (Participants) | 9 | 13 | 7
  Day 17/predose | 63.94 (8.928) | 67.46 (7.148) | 72.49 (6.267)
  Day 17/2h postdose: number analyzed (Participants) | 9 | 13 | 6
  Day 17/2h postdose | 69.37 (13.141) | 71.81 (7.052) | 79.18 (10.040)
  Day 17/4h postdose: number analyzed (Participants) | 9 | 13 | 6
  Day 17/4h postdose | 65.22 (11.339) | 67.85 (6.367) | 72.80 (8.155)
  Day 17/8h postdose: number analyzed (Participants) | 9 | 13 | 6
  Day 17/8h postdose | 65.33 (10.546) | 69.58 (9.254) | 75.43 (6.394)
  Day 17/12h postdose: number analyzed (Participants) | 9 | 13 | 6
  Day 17/12h postdose | 72.99 (13.349) | 73.61 (6.739) | 84.45 (13.229)
  Day 20/predose: number analyzed (Participants) | 9 | 13 | 5
  Day 20/predose | 65.01 (8.519) | 67.86 (7.128) | 75.48 (12.388)
  Day 20/2h postdose: number analyzed (Participants) | 9 | 13 | 5
  Day 20/2h postdose | 71.04 (11.835) | 75.92 (7.602) | 77.66 (9.390)
  Day 20/4h postdose: number analyzed (Participants) | 9 | 13 | 5
  Day 20/4h postdose | 65.81 (9.536) | 71.79 (8.061) | 73.86 (9.380)
  Day 20/8h postdose: number analyzed (Participants) | 9 | 13 | 5
  Day 20/8h postdose | 64.78 (8.599) | 71.41 (7.260) | 74.08 (10.559)
  Day 20/12h postdose: number analyzed (Participants) | 9 | 13 | 5
  Day 20/12h postdose | 72.33 (11.407) | 76.69 (8.385) | 81.60 (12.056)
  Day 23/predose: number analyzed (Participants) | 9 | 12 | 5
  Day 23/predose | 63.14 (10.228) | 71.69 (11.467) | 75.68 (8.004)
  Day 23/2h postdose: number analyzed (Participants) | 9 | 12 | 5
  Day 23/2h postdose | 71.97 (14.111) | 77.33 (8.980) | 78.92 (5.821)
  Day 23/4h postdose: number analyzed (Participants) | 9 | 12 | 5
  Day 23/4h postdose | 68.33 (14.452) | 73.53 (12.354) | 73.90 (8.044)
  Day 23/8h postdose: number analyzed (Participants) | 9 | 12 | 5
  Day 23/8h postdose | 68.04 (14.294) | 73.88 (10.252) | 74.28 (4.754)
  Day 23/12h postdose: number analyzed (Participants) | 9 | 12 | 5
  Day 23/12h postdose | 75.03 (12.274) | 77.75 (10.730) | 82.00 (9.300)
  Day 15/predose (metop. 25 mg): number analyzed (Participants) | 3 | 4 | 3
  Day 15/predose (metop. 25 mg) | 64.03 (7.024) | 59.48 (2.873) | 73.67 (5.677)
  Day 15/2h postdose (metop. 25 mg): number analyzed (Participants) | 3 | 4 | 3
  Day 15/2h postdose (metop. 25 mg) | 72.13 (13.967) | 63.18 (3.767) | 78.77 (3.044)
  Day 15/4h postdose (metop. 25 mg): number analyzed (Participants) | 3 | 4 | 3
  Day 15/4h postdose (metop. 25 mg) | 63.87 (11.356) | 55.73 (4.057) | 71.90 (3.483)
  Day 15/8h postdose (metop. 25 mg): number analyzed (Participants) | 3 | 4 | 3
  Day 15/8h postdose (metop. 25 mg) | 63.67 (11.257) | 58.23 (1.776) | 73.10 (7.045)
  Day 15/12h postdose (metop. 25 mg): number analyzed (Participants) | 3 | 4 | 3
  Day 15/12h postdose (metop. 25 mg) | 64.23 (15.989) | 60.85 (4.615) | 79.53 (7.012)
  Day 18/predose (metop. 25 mg): number analyzed (Participants) | 5 | 5 | 2
  Day 18/predose (metop. 25 mg) | 62.28 (7.486) | 71.40 (9.612) | 97.20 (27.577)
  Day 18/2h postdose (metop. 25 mg): number analyzed (Participants) | 5 | 5 | 2
  Day 18/2h postdose (metop. 25 mg) | 65.82 (7.663) | 71.78 (4.462) | 83.65 (10.819)
  Day 18/4h postdose (metop. 25 mg): number analyzed (Participants) | 5 | 5 | 2
  Day 18/4h postdose (metop. 25 mg) | 57.72 (4.800) | 69.40 (6.557) | 80.50 (14.425)
  Day 18/8h postdose (metop. 25 mg): number analyzed (Participants) | 5 | 5 | 2
  Day 18/8h postdose (metop. 25 mg) | 59.34 (4.298) | 73.14 (8.564) | 82.85 (12.516)
  Day 18/12h postdose (metop. 25 mg): number analyzed (Participants) | 5 | 5 | 2
  Day 18/12h postdose (metop. 25 mg) | 62.34 (5.816) | 76.80 (8.243) | 87.00 (6.081)
  Day 21/predose (metop. 25 mg): number analyzed (Participants) | 1 | 4 | 1
  Day 21/predose (metop. 25 mg) | 73.30 (NA) — NA=not calculated/1 subject | 76.90 (3.344) | 72.00 (NA) — NA=not calculated/1 subject
  Day 21/2h postdose (metop. 25 mg): number analyzed (Participants) | 1 | 4 | 1
  Day 21/2h postdose (metop. 25 mg) | 75.70 (NA) — NA=not calculated/1 subject | 80.00 (5.170) | 68.70 (NA) — NA=not calculated/1 subject
  Day 21/4h postdose (metop. 25 mg): number analyzed (Participants) | 1 | 4 | 1
  Day 21/4h postdose (metop. 25 mg) | 77.00 (NA) — NA=not calculated/1 subject | 73.23 (2.165) | 70.70 (NA) — NA=not calculated/1 subject
  Day 21/8h postdose (metop. 25 mg): number analyzed (Participants) | 1 | 4 | 1
  Day 21/8h postdose (metop. 25 mg) | 72.70 (NA) — NA=not calculated/1 subject | 71.40 (4.723) | 64.00 (NA) — NA=not calculated/1 subject
  Day 21/12h postdose (metop. 25 mg): number analyzed (Participants) | 1 | 4 | 1
  Day 21/12h postdose (metop. 25 mg) | 80.0 (NA) — NA=not calculated/1 subject | 74.23 (3.015) | 74.70 (NA) — NA=not calculated/1 subject
  Day 15/predose (metop. 50 mg): number analyzed (Participants) | 3 | 3 | 2
  Day 15/predose (metop. 50 mg) | 61.43 (10.112) | 70.47 (6.353) | 74.85 (0.212)
  Day 15/2h postdose (metop. 50 mg): number analyzed (Participants) | 3 | 3 | 2
  Day 15/2h postdose (metop. 50 mg) | 65.10 (9.986) | 74.00 (5.568) | 75.15 (6.859)
  Day 15/4h postdose (metop. 50 mg): number analyzed (Participants) | 3 | 3 | 2
  Day 15/4h postdose (metop. 50 mg) | 60.43 (10.327) | 67.47 (4.895) | 70.85 (0.212)
  Day 15/8h postdose (metop. 50 mg): number analyzed (Participants) | 3 | 3 | 2
  Day 15/8h postdose (metop. 50 mg) | 59.67 (9.205) | 69.10 (7.136) | 66.70 (1.414)
  Day 15/12h postdose (metop. 50 mg): number analyzed (Participants) | 3 | 3 | 2
  Day 15/12h postdose (metop. 50 mg) | 65.00 (9.853) | 74.33 (3.953) | 71.20 (4.950)
  Day 18/predose (metop. 50 mg): number analyzed (Participants) | 3 | 6 | 1
  Day 18/predose (metop. 50 mg) | 66.00 (13.454) | 67.17 (7.909) | 88.70 (NA) — NA=not calculated/1 subject
  Day 18/2h postdose (metop. 50 mg): number analyzed (Participants) | 3 | 6 | 1
  Day 18/2h postdose (metop. 50 mg) | 72.13 (16.783) | 71.72 (7.843) | 100.00 (NA) — NA=not calculated/1 subject
  Day 18/4h postdose (metop. 50 mg): number analyzed (Participants) | 3 | 6 | 1
  Day 18/4h postdose (metop. 50 mg) | 62.57 (12.307) | 64.50 (7.223) | 90.30 (NA) — NA=not calculated/1 subject
  Day 18/8h postdose (metop. 50 mg): number analyzed (Participants) | 3 | 6 | 1
  Day 18/8h postdose (metop. 50 mg) | 63.10 (14.509) | 61.88 (6.462) | 79.70 (NA) — NA=not calculated/1 subject
  Day 18/12h postdose (metop. 50 mg): number analyzed (Participants) | 3 | 6 | 1
  Day 18/12h postdose (metop. 50 mg) | 65.70 (14.526) | 64.38 (6.019) | 86.30 (NA) — NA=not calculated/1 subject
  Day 21/predose (metop. 50 mg): number analyzed (Participants) | 3 | 4 | 3
  Day 21/predose (metop. 50 mg) | 63.53 (2.658) | 65.25 (7.722) | 81.67 (16.359)
  Day 21/2h postdose (metop. 50 mg): number analyzed (Participants) | 3 | 4 | 3
  Day 21/2h postdose (metop. 50 mg) | 64.90 (5.188) | 71.33 (13.126) | 79.20 (10.613)
  Day 21/4h postdose (metop. 50 mg): number analyzed (Participants) | 3 | 4 | 3
  Day 21/4h postdose (metop. 50 mg) | 60.90 (9.106) | 64.75 (8.048) | 71.67 (10.855)
  Day 21/8h postdose (metop. 50 mg): number analyzed (Participants) | 3 | 4 | 3
  Day 21/8h postdose (metop. 50 mg) | 61.97 (15.144) | 62.83 (6.737) | 74.33 (6.987)
  Day 21/12h postdose (metop. 50 mg): number analyzed (Participants) | 3 | 4 | 3
  Day 21/12h postdose (metop. 50 mg) | 61.33 (4.384) | 67.00 (8.922) | 78.13 (8.790)
  Day 15/predose (metop. 100 mg): number analyzed (Participants) | 3 | 6 | 2
  Day 15/predose (metop. 100 mg) | 70.00 (6.324) | 68.83 (5.611) | 79.50 (17.253)
  Day 15/2h postdose (metop. 100 mg): number analyzed (Participants) | 3 | 6 | 2
  Day 15/2h postdose (metop. 100 mg) | 60.70 (3.000) | 68.28 (3.520) | 68.15 (8.697)
  Day 15/4h postdose (metop. 100 mg): number analyzed (Participants) | 3 | 6 | 2
  Day 15/4h postdose (metop. 100 mg) | 54.53 (1.079) | 59.97 (3.989) | 65.80 (7.778)
  Day 15/8h postdose (metop. 100 mg): number analyzed (Participants) | 3 | 6 | 2
  Day 15/8h postdose (metop. 100 mg) | 56.57 (6.772) | 61.88 (10.818) | 65.15 (6.859)
  Day 15/12h postdose (metop. 100 mg): number analyzed (Participants) | 3 | 6 | 2
  Day 15/12h postdose (metop. 100 mg) | 56.57 (0.513) | 65.18 (6.649) | 71.50 (10.182)
  Day 18/predose (metop. 100 mg): number analyzed (Participants) | 1 | 2 | 3
  Day 18/predose (metop. 100 mg) | 72.00 (NA) — NA=not calculated/1 subject | 68.35 (10.394) | 73.74 (3.356)
  Day 18/2h postdose (metop. 100 mg): number analyzed (Participants) | 1 | 2 | 3
  Day 18/2h postdose (metop. 100 mg) | 76.70 (NA) — NA=not calculated/1 subject | 65.65 (9.405) | 74.33 (8.736)
  Day 18/4h postdose (metop. 100 mg): number analyzed (Participants) | 1 | 2 | 3
  Day 18/4h postdose (metop. 100 mg) | 70.0 (NA) — NA=not calculated/1 subject | 61.00 (8.061) | 66.10 (10.198)
  Day 18/8h postdose (metop. 100 mg): number analyzed (Participants) | 1 | 2 | 3
  Day 18/8h postdose (metop. 100 mg) | 72.30 (NA) — NA=not calculated/1 subject | 58.35 (8.980) | 65.23 (3.233)
  Day 18/12h postdose (metop. 100 mg): number analyzed (Participants) | 1 | 2 | 3
  Day 18/12h postdose (metop. 100 mg) | 77.30 (NA) — NA=not calculated/1 subject | 62.30 (2.828) | 71.33 (9.292)
  Day 21/predose (metop. 100 mg): number analyzed (Participants) | 5 | 5 | 1
  Day 21/predose (metop. 100 mg) | 64.60 (11.603) | 67.08 (8.499) | 76.00 (NA) — NA=not calculated/1 subject
  Day 21/2h postdose (metop. 100 mg): number analyzed (Participants) | 5 | 5 | 1
  Day 21/2h postdose (metop. 100 mg) | 69.14 (14.391) | 69.66 (11.330) | 63.70 (NA) — NA=not calculated/1 subject
  Day 21/4h postdose (metop. 100 mg): number analyzed (Participants) | 5 | 5 | 1
  Day 21/4h postdose (metop. 100 mg) | 60.12 (11.471) | 60.66 (9.142) | 56.00 (NA) — NA=not calculated/1 subject
  Day 21/8h postdose (metop. 100 mg): number analyzed (Participants) | 5 | 5 | 1
  Day 21/8h postdose (metop. 100 mg) | 59.72 (11.113) | 61.66 (11.039) | 56.70 (NA) — NA=not calculated/1 subject
  Day 21/12h postdose (metop. 100 mg): number analyzed (Participants) | 5 | 5 | 1
  Day 21/12h postdose (metop. 100 mg) | 65.34 (13.190) | 68.06 (9.870) | 71.70 (NA) — NA=not calculated/1 subject

11. Secondary Outcome: Diastolic Blood Pressure (DBP) and Systolic Blood Pressure (SBP) Values After at Least 10 Minutes Rest Before Each PK Sampling Time Point or the Corresponding Time Point (Day -1, Day 13 [Pre-dose Only], Day 14, 15, 17, 18, 20, 21, 23)
Time Frame: Day -1, Day 13 [pre-dose only], Day 14, Day 15, Day 17, Day 18, Day 20, Day 21 and Day 23
Population: All subjects included in the study and dosed with IMP were included in the safety population. The number of participants listed below is the number of subjects with an assessment at the specified time point.
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Cohort 1 (Tesofensine 0.25mg) | Cohort 2 (Tesofensine 0.50mg) | Cohort 3 (Tesofensine 0.75mg)
Number analyzed (Participants) | 9 | 16 | 12
mm Hg
  DBP Day -1/predose | 73.09 (8.953) | 71.00 (5.235) | 73.83 (5.838)
  DBP Day -1/2h postdose | 67.07 (7.998) | 63.87 (7.387) | 69.66 (5.233)
  DBP Day -1/4h postdose | 70.26 (9.593) | 68.68 (4.609) | 71.86 (5.184)
  DBP Day -1/8h postdose | 72.11 (9.712) | 69.39 (5.265) | 74.88 (5.346)
  DBP Day -1/12h postdose | 68.91 (9.942) | 66.66 (5.051) | 71.27 (6.221)
  DBP Day 13/predose: number analyzed (Participants) | 9 | 14 | 7
  DBP Day 13/predose | 70.48 (10.740) | 71.24 (5.017) | 77.79 (7.288)
  DBP Day 14/predose: number analyzed (Participants) | 9 | 14 | 7
  DBP Day 14/predose | 71.16 (10.810) | 71.58 (6.727) | 77.73 (5.384)
  DBP Day 14/2h postdose: number analyzed (Participants) | 9 | 14 | 7
  DBP Day 14/2h postdose | 68.94 (9.394) | 67.23 (5.930) | 75.13 (7.129)
  DBP Day 14/4h postdose: number analyzed (Participants) | 9 | 14 | 7
  DBP Day 14/4h postdose | 71.00 (8.895) | 70.19 (5.499) | 77.54 (7.374)
  DBP Day 14/8h postdose: number analyzed (Participants) | 9 | 14 | 7
  DBP Day 14/8h postdose | 74.08 (10.285) | 72.23 (6.881) | 77.49 (4.556)
  DBP Day 14/12h postdose: number analyzed (Participants) | 9 | 14 | 7
  DBP Day 14/12h postdose | 73.12 (8.227) | 70.08 (6.681) | 76.69 (5.087)
  DBP Day 17/predose: number analyzed (Participants) | 9 | 13 | 7
  DBP Day 17/predose | 70.68 (9.731) | 70.76 (4.939) | 75.90 (5.160)
  DBP Day 17/2h postdose: number analyzed (Participants) | 9 | 13 | 6
  DBP Day 17/2h postdose | 68.70 (10.010) | 67.91 (5.120) | 75.83 (5.199)
  DBP Day 17/4h postdose: number analyzed (Participants) | 9 | 13 | 6
  DBP Day 17/4h postdose | 70.11 (9.157) | 70.75 (5.893) | 78.65 (8.054)
  DBP Day 17/8h postdose: number analyzed (Participants) | 9 | 13 | 6
  DBP Day 17/8h postdose | 70.96 (9.215) | 70.97 (7.122) | 81.38 (7.746)
  DBP Day 17/12h postdose: number analyzed (Participants) | 9 | 13 | 6
  DBP Day 17/12h postdose | 70.89 (9.080) | 70.15 (6.363) | 78.38 (8.679)
  DBP Day 20/predose: number analyzed (Participants) | 9 | 13 | 5
  DBP Day 20/predose | 71.12 (10.779) | 68.89 (6.413) | 75.08 (9.153)
  DBP Day 20/2h postdose: number analyzed (Participants) | 9 | 13 | 5
  DBP Day 20/2h postdose | 68.70 (7.133) | 67.54 (4.643) | 75.48 (11.316)
  DBP Day 20/4h postdose: number analyzed (Participants) | 9 | 13 | 5
  DBP Day 20/4h postdose | 69.88 (8.037) | 69.85 (5.340) | 78.08 (7.286)
  DBP Day 20/8h postdose: number analyzed (Participants) | 9 | 13 | 5
  DBP Day 20/8h postdose | 72.27 (8.309) | 71.18 (6.024) | 77.80 (9.539)
  DBP Day 20/12h postdose: number analyzed (Participants) | 9 | 13 | 5
  DBP Day 20/12h postdose | 70.38 (9.396) | 69.99 (4.541) | 76.14 (9.077)
  DBP Day 23/predose: number analyzed (Participants) | 9 | 12 | 5
  DBP Day 23/predose | 69.46 (10.420) | 71.55 (6.831) | 78.88 (3.275)
  DBP Day 23/2h postdose: number analyzed (Participants) | 9 | 12 | 5
  DBP Day 23/2h postdose | 66.19 (8.480) | 68.50 (6.328) | 77.54 (8.795)
  DBP Day 23/4h postdose: number analyzed (Participants) | 9 | 12 | 5
  DBP Day 23/4h postdose | 70.49 (9.973) | 71.54 (7.256) | 81.34 (6.330)
  DBP Day 23/8h postdose: number analyzed (Participants) | 9 | 12 | 5
  DBP Day 23/8h postdose | 72.13 (8.899) | 74.52 (7.792) | 82.26 (7.506)
  DBP Day 23/12h postdose: number analyzed (Participants) | 9 | 12 | 5
  DBP Day 23/12h postdose | 70.92 (8.500) | 73.93 (6.405) | 81.14 (6.935)
  DBP Day 15/predose (metop. 25 mg): number analyzed (Participants) | 3 | 4 | 3
  DBP Day 15/predose (metop. 25 mg) | 77.47 (7.257) | 74.25 (3.817) | 79.90 (4.257)
  DBP Day 15/2h postdose (metop. 25 mg): number analyzed (Participants) | 3 | 4 | 3
  DBP Day 15/2h postdose (metop. 25 mg) | 76.53 (7.594) | 67.78 (4.541) | 76.67 (5.677)
  DBP Day 15/4h postdose (metop. 25 mg): number analyzed (Participants) | 3 | 4 | 3
  DBP Day 15/4h postdose (metop. 25 mg) | 81.00 (7.000) | 72.68 (5.068) | 75.20 (5.327)
  DBP Day 15/8h postdose (metop. 25 mg): number analyzed (Participants) | 3 | 4 | 3
  DBP Day 15/8h postdose (metop. 25 mg) | 78.20 (8.940) | 73.00 (6.947) | 78.33 (6.207)
  DBP Day 15/12h postdose (metop. 25 mg): number analyzed (Participants) | 3 | 4 | 3
  DBP Day 15/12h postdose (metop. 25 mg) | 77.10 (7.970) | 70.58 (3.837) | 74.00 (5.205)
  DBP Day 18/predose (metop. 25 mg): number analyzed (Participants) | 5 | 5 | 2
  DBP Day 18/predose (metop. 25 mg) | 69.34 (6.846) | 71.60 (8.405) | 83.50 (17.678)
  DBP Day 18/2h postdose (metop. 25 mg): number analyzed (Participants) | 5 | 5 | 2
  DBP Day 18/2h postdose (metop. 25 mg) | 66.74 (6.906) | 68.28 (7.602) | 77.85 (14.354)
  DBP Day 18/4h postdose (metop. 25 mg): number analyzed (Participants) | 5 | 5 | 2
  DBP Day 18/4h postdose (metop. 25 mg) | 66.80 (9.121) | 69.16 (8.603) | 78.20 (12.021)
  DBP Day 18/8h postdose (metop. 25 mg): number analyzed (Participants) | 5 | 5 | 2
  DBP Day 18/8h postdose (metop. 25 mg) | 68.52 (7.826) | 69.54 (10.062) | 78.00 (15.981)
  DBP Day 18/12h postdose (metop. 25 mg): number analyzed (Participants) | 5 | 5 | 2
  DBP Day 18/12h postdose (metop. 25 mg) | 67.58 (7.949) | 69.26 (7.755) | 78.15 (13.930)
  DBP Day 21/predose (metop. 25 mg): number analyzed (Participants) | 1 | 4 | 1
  DBP Day 21/predose (metop. 25 mg) | 65.70 (NA) — NA=not calculated/1 subject | 73.40 (2.859) | 82.70 (NA) — NA=not calculated/1 subject
  DBP Day 21/2h postdose (metop. 25 mg): number analyzed (Participants) | 1 | 4 | 1
  DBP Day 21/2h postdose (metop. 25 mg) | 65.00 (NA) — NA=not calculated/1 subject | 70.35 (4.159) | 77.30 (NA) — NA=not calculated/1 subject
  DBP Day 21/4h postdose (metop. 25 mg): number analyzed (Participants) | 1 | 4 | 1
  DBP Day 21/4h postdose (metop. 25 mg) | 64.70 (NA) — NA=not calculated/1 subject | 70.93 (5.734) | 81.70 (NA) — NA=not calculated/1 subject
  DBP Day 21/8h postdose (metop. 25 mg): number analyzed (Participants) | 1 | 4 | 1
  DBP Day 21/8h postdose (metop. 25 mg) | 65.70 (NA) — NA=not calculated/1 subject | 73.60 (6.902) | 75.70 (NA) — NA=not calculated/1 subject
  DBP Day 21/12h postdose (metop. 25 mg): number analyzed (Participants) | 1 | 4 | 1
  DBP Day 21/12h postdose (metop. 25 mg) | 62.70 (NA) — NA=not calculated/1 subject | 71.15 (7.964) | 81.00 (NA) — NA=not calculated/1 subject
  DBP Day 15/predose (metop. 50 mg): number analyzed (Participants) | 3 | 3 | 2
  DBP Day 15/predose (metop. 50 mg) | 73.90 (7.016) | 78.33 (10.795) | 77.50 (9.617)
  DBP Day 15/2h postdose (metop. 50 mg): number analyzed (Participants) | 3 | 3 | 2
  DBP Day 15/2h postdose (metop. 50 mg) | 67.00 (1.179) | 71.87 (7.467) | 73.50 (12.445)
  DBP Day 15/4h postdose (metop. 50 mg): number analyzed (Participants) | 3 | 3 | 2
  DBP Day 15/4h postdose (metop. 50 mg) | 72.23 (4.761) | 73.00 (6.032) | 74.80 (10.607)
  DBP Day 15/8h postdose (metop. 50 mg): number analyzed (Participants) | 3 | 3 | 2
  DBP Day 15/8h postdose (metop. 50 mg) | 67.90 (6.537) | 72.57 (10.657) | 71.50 (4.525)
  DBP Day 15/12h postdose (metop. 50 mg): number analyzed (Participants) | 3 | 3 | 2
  DBP Day 15/12h postdose (metop. 50 mg) | 70.00 (7.550) | 74.20 (6.183) | 69.50 (1.131)
  DBP Day 18/predose (metop. 50 mg): number analyzed (Participants) | 3 | 6 | 1
  DBP Day 18/predose (metop. 50 mg) | 80.47 (8.495) | 71.83 (5.043) | 80.00 (NA) — NA=not calculated/1 subject
  DBP Day 18/2h postdose (metop. 50 mg): number analyzed (Participants) | 3 | 6 | 1
  DBP Day 18/2h postdose (metop. 50 mg) | 74.23 (4.225) | 65.95 (3.651) | 80.30 (NA) — NA=not calculated/1 subject
  DBP Day 18/4h postdose (metop. 50 mg): number analyzed (Participants) | 3 | 6 | 1
  DBP Day 18/4h postdose (metop. 50 mg) | 75.97 (5.033) | 69.05 (7.023) | 82.00 (NA) — NA=not calculated/1 subject
  DBP Day 18/8h postdose (metop. 50 mg): number analyzed (Participants) | 3 | 6 | 1
  DBP Day 18/8h postdose (metop. 50 mg) | 79.77 (9.474) | 73.33 (4.235) | 80.70 (NA) — NA=not calculated/1 subject
  DBP Day 18/12h postdose (metop. 50 mg): number analyzed (Participants) | 3 | 6 | 1
  DBP Day 18/12h postdose (metop. 50 mg) | 74.23 (6.933) | 66.82 (4.704) | 80.70 (NA) — NA=not calculated/1 subject
  DBP Day 21/predose (metop. 50 mg): number analyzed (Participants) | 3 | 4 | 3
  DBP Day 21/predose (metop. 50 mg) | 65.00 (11.287) | 68.58 (5.169) | 83.90 (10.523)
  DBP Day 21/2h postdose (metop. 50 mg): number analyzed (Participants) | 3 | 4 | 3
  DBP Day 21/2h postdose (metop. 50 mg) | 61.67 (12.314) | 65.08 (3.428) | 80.10 (9.226)
  DBP Day 21/4h postdose (metop. 50 mg): number analyzed (Participants) | 3 | 4 | 3
  DBP Day 21/4h postdose (metop. 50 mg) | 63.67 (10.365) | 66.68 (4.261) | 82.10 (10.860)
  DBP Day 21/8h postdose (metop. 50 mg): number analyzed (Participants) | 3 | 4 | 3
  DBP Day 21/8h postdose (metop. 50 mg) | 66.43 (1.401) | 65.83 (6.081) | 79.00 (9.154)
  DBP Day 21/12h postdose (metop. 50 mg): number analyzed (Participants) | 3 | 4 | 3
  DBP Day 21/12h postdose (metop. 50 mg) | 61.67 (6.747) | 66.08 (3.175) | 75.13 (9.152)
  DBP Day 15/predose (metop. 100 mg): number analyzed (Participants) | 3 | 6 | 2
  DBP Day 15/predose (metop. 100 mg) | 67.43 (9.125) | 69.95 (4.216) | 85.00 (12.304)
  DBP Day 15/2h postdose (metop. 100 mg): number analyzed (Participants) | 3 | 6 | 2
  DBP Day 15/2h postdose (metop. 100 mg) | 62.80 (10.641) | 63.73 (3.037) | 78.00 (11.314)
  DBP Day 15/4h postdose (metop. 100 mg): number analyzed (Participants) | 3 | 6 | 2
  DBP Day 15/4h postdose (metop. 100 mg) | 59.13 (10.304) | 67.78 (5.407) | 79.00 (6.647)
  DBP Day 15/8h postdose (metop. 100 mg): number analyzed (Participants) | 3 | 6 | 2
  DBP Day 15/8h postdose (metop. 100 mg) | 62.57 (5.954) | 67.10 (5.255) | 82.85 (4.455)
  DBP Day 15/12h postdose (metop. 100 mg): number analyzed (Participants) | 3 | 6 | 2
  DBP Day 15/12h postdose (metop. 100 mg) | 58.47 (11.898) | 64.67 (5.343) | 77.00 (3.818)
  DBP Day 18/predose (metop. 100 mg): number analyzed (Participants) | 1 | 2 | 3
  DBP Day 18/predose (metop. 100 mg) | 67.00 (NA) — NA=not calculated/1 subject | 75.30 (1.414) | 78.57 (1.858)
  DBP Day 18/2h postdose (metop. 100 mg): number analyzed (Participants) | 1 | 2 | 3
  DBP Day 18/2h postdose (metop. 100 mg) | 62.70 (NA) — NA=not calculated/1 subject | 74.65 (1.909) | 75.10 (5.303)
  DBP Day 18/4h postdose (metop. 100 mg): number analyzed (Participants) | 1 | 2 | 3
  DBP Day 18/4h postdose (metop. 100 mg) | 68.30 (NA) — NA=not calculated/1 subject | 76.00 (4.667) | 75.57 (5.353)
  DBP Day 18/8h postdose (metop. 100 mg): number analyzed (Participants) | 1 | 2 | 3
  DBP Day 18/8h postdose (metop. 100 mg) | 65.00 (NA) — NA=not calculated/1 subject | 69.65 (0.495) | 77.90 (3.305)
  DBP Day 18/12h postdose (metop. 100 mg): number analyzed (Participants) | 1 | 2 | 3
  DBP Day 18/12h postdose (metop. 100 mg) | 63.00 (NA) — NA=not calculated/1 subject | 72.00 (2.404) | 73.10 (3.568)
  DBP Day 21/predose (metop. 100 mg): number analyzed (Participants) | 5 | 5 | 1
  DBP Day 21/predose (metop. 100 mg) | 75.08 (8.627) | 73.62 (6.640) | 71.30 (NA) — NA=not calculated/1 subject
  DBP Day 21/2h postdose (metop. 100 mg): number analyzed (Participants) | 5 | 5 | 1
  DBP Day 21/2h postdose (metop. 100 mg) | 72.60 (6.741) | 69.14 (4.944) | 68.70 (NA) — NA=not calculated/1 subject
  DBP Day 21/4h postdose (metop. 100 mg): number analyzed (Participants) | 5 | 5 | 1
  DBP Day 21/4h postdose (metop. 100 mg) | 75.52 (6.615) | 72.60 (5.019) | 72.70 (NA) — NA=not calculated/1 subject
  DBP Day 21/8h postdose (metop. 100 mg): number analyzed (Participants) | 5 | 5 | 1
  DBP Day 21/8h postdose (metop. 100 mg) | 75.86 (6.464) | 72.80 (4.727) | 74.70 (NA) — NA=not calculated/1 subject
  DBP Day 21/12h postdose (metop. 100 mg): number analyzed (Participants) | 5 | 5 | 1
  DBP Day 21/12h postdose (metop. 100 mg) | 72.06 (5.056) | 71.86 (3.734) | 71.70 (NA) — NA=not calculated/1 subject
  SBP Day -1/predose | 116.30 (8.897) | 113.51 (6.626) | 119.97 (7.666)
  SBP Day -1/2h postdose | 113.40 (4.560) | 108.13 (9.565) | 116.34 (7.740)
  SBP Day -1/4h postdose | 115.03 (12.772) | 112.65 (10.492) | 118.01 (9.510)
  SBP Day -1/8h postdose | 117.87 (10.346) | 114.22 (8.844) | 123.13 (10.019)
  SBP Day -1/12h postdose | 118.97 (11.269) | 112.79 (11.262) | 119.76 (9.957)
  SBP Day 13/predose: number analyzed (Participants) | 9 | 14 | 7
  SBP Day 13/predose | 116.26 (12.894) | 116.44 (10.639) | 123.29 (13.645)
  SBP Day 14/predose: number analyzed (Participants) | 9 | 14 | 7
  SBP Day 14/predose | 116.79 (11.931) | 115.53 (11.630) | 123.33 (13.602)
  SBP Day 14/2h postdose: number analyzed (Participants) | 9 | 14 | 7
  SBP Day 14/2h postdose | 117.11 (10.406) | 111.74 (10.479) | 124.29 (14.259)
  SBP Day 14/4h postdose: number analyzed (Participants) | 9 | 14 | 7
  SBP Day 14/4h postdose | 118.73 (9.790) | 116.83 (9.799) | 125.94 (12.902)
  SBP Day 14/8h postdose: number analyzed (Participants) | 9 | 14 | 7
  SBP Day 14/8h postdose | 121.03 (11.850) | 118.69 (12.810) | 125.01 (13.571)
  SBP Day 14/12h postdose: number analyzed (Participants) | 9 | 14 | 7
  SBP Day 14/12h postdose | 121.37 (12.372) | 117.85 (12.695) | 124.34 (14.504)
  SBP Day 17/predose: number analyzed (Participants) | 9 | 13 | 7
  SBP Day 17/predose | 113.40 (12.694) | 115.64 (9.746) | 124.71 (10.037)
  SBP Day 17/2h postdose: number analyzed (Participants) | 9 | 13 | 6
  SBP Day 17/2h postdose | 115.81 (12.775) | 112.82 (10.935) | 122.77 (10.881)
  SBP Day 17/4h postdose: number analyzed (Participants) | 9 | 13 | 6
  SBP Day 17/4h postdose | 118.51 (11.659) | 117.53 (10.373) | 125.48 (11.657)
  SBP Day 17/8h postdose: number analyzed (Participants) | 9 | 13 | 6
  SBP Day 17/8h postdose | 118.60 (14.297) | 119.01 (11.850) | 129.22 (13.063)
  SBP Day 17/12h postdose: number analyzed (Participants) | 9 | 13 | 6
  SBP Day 17/12h postdose | 121.37 (14.208) | 120.24 (12.660) | 131.12 (15.701)
  SBP Day 20/predose: number analyzed (Participants) | 9 | 13 | 5
  SBP Day 20/predose | 116.07 (12.769) | 113.80 (11.463) | 122.52 (16.577)
  SBP Day 20/2h postdose: number analyzed (Participants) | 9 | 13 | 5
  SBP Day 20/2h postdose | 114.89 (13.293) | 113.92 (11.205) | 126.00 (11.011)
  SBP Day 20/4h postdose: number analyzed (Participants) | 9 | 13 | 5
  SBP Day 20/4h postdose | 118.20 (11.076) | 114.44 (10.849) | 128.54 (13.331)
  SBP Day 20/8h postdose: number analyzed (Participants) | 9 | 13 | 5
  SBP Day 20/8h postdose | 120.89 (11.552) | 117.78 (12.058) | 127.28 (16.690)
  SBP Day 20/12h postdose: number analyzed (Participants) | 9 | 13 | 5
  SBP Day 20/12h postdose | 119.97 (13.690) | 116.58 (10.778) | 128.62 (11.530)
  SBP Day 23/predose: number analyzed (Participants) | 9 | 12 | 5
  SBP Day 23/predose | 114.92 (14.228) | 116.43 (13.179) | 126.46 (7.896)
  SBP Day 23/2h postdose: number analyzed (Participants) | 9 | 12 | 5
  SBP Day 23/2h postdose | 111.79 (12.343) | 113.05 (12.730) | 126.46 (12.526)
  SBP Day 23/4h postdose: number analyzed (Participants) | 9 | 12 | 5
  SBP Day 23/4h postdose | 118.07 (11.363) | 117.38 (13.244) | 130.40 (9.270)
  SBP Day 23/8h postdose: number analyzed (Participants) | 9 | 12 | 5
  SBP Day 23/8h postdose | 117.46 (12.443) | 121.24 (14.711) | 130.00 (11.933)
  SBP Day 23/12h postdose: number analyzed (Participants) | 9 | 12 | 5
  SBP Day 23/12h postdose | 121.09 (12.568) | 124.08 (14.322) | 131.80 (10.082)
  SBP Day 15/predose (metop. 25 mg): number analyzed (Participants) | 3 | 4 | 3
  SBP Day 15/predose (metop. 25 mg) | 121.67 (7.343) | 118.80 (5.916) | 120.90 (2.476)
  SBP Day 15/2h postdose (metop. 25 mg): number analyzed (Participants) | 3 | 4 | 3
  SBP Day 15/2h postdose (metop. 25 mg) | 122.80 (11.177) | 111.50 (6.104) | 121.67 (4.245)
  SBP Day 15/4h postdose (metop. 25 mg): number analyzed (Participants) | 3 | 4 | 3
  SBP Day 15/4h postdose (metop. 25 mg) | 124.67 (13.683) | 117.43 (6.098) | 117.30 (1.000)
  SBP Day 15/8h postdose (metop. 25 mg): number analyzed (Participants) | 3 | 4 | 3
  SBP Day 15/8h postdose (metop. 25 mg) | 124.80 (12.909) | 124.35 (13.169) | 124.23 (5.437)
  SBP Day 15/12h postdose (metop. 25 mg): number analyzed (Participants) | 3 | 4 | 3
  SBP Day 15/12h postdose (metop. 25 mg) | 126.33 (10.398) | 119.33 (9.947) | 121.10 (5.986)
  SBP Day 18/predose (metop. 25 mg): number analyzed (Participants) | 5 | 5 | 2
  SBP Day 18/predose (metop. 25 mg) | 113.14 (9.615) | 114.26 (13.264) | 141.35 (38.679)
  SBP Day 18/2h postdose (metop. 25 mg): number analyzed (Participants) | 5 | 5 | 2
  SBP Day 18/2h postdose (metop. 25 mg) | 115.14 (10.768) | 109.66 (12.729) | 127.00 (25.032)
  SBP Day 18/4h postdose (metop. 25 mg): number analyzed (Participants) | 5 | 5 | 2
  SBP Day 18/4h postdose (metop. 25 mg) | 114.46 (12.510) | 112.60 (15.101) | 130.20 (20.506)
  SBP Day 18/8h postdose (metop. 25 mg): number analyzed (Participants) | 5 | 5 | 2
  SBP Day 18/8h postdose (metop. 25 mg) | 118.72 (11.574) | 112.88 (14.848) | 133.00 (29.274)
  SBP Day 18/12h postdose (metop. 25 mg): number analyzed (Participants) | 5 | 5 | 2
  SBP Day 18/12h postdose (metop. 25 mg) | 118.02 (15.047) | 113.74 (15.735) | 134.35 (24.537)
  SBP Day 21/predose (metop. 25 mg): number analyzed (Participants) | 1 | 4 | 1
  SBP Day 21/predose (metop. 25 mg) | 108.70 (NA) — NA=not calculated/1 subject | 123.15 (16.418) | 139.70 (NA) — NA=not calculated/1 subject
  SBP Day 21/2h postdose (metop. 25 mg): number analyzed (Participants) | 1 | 4 | 1
  SBP Day 21/2h postdose (metop. 25 mg) | 116.70 (NA) — NA=not calculated/1 subject | 115.83 (11.601) | 133.00 (NA) — NA=not calculated/1 subject
  SBP Day 21/4h postdose (metop. 25 mg): number analyzed (Participants) | 1 | 4 | 1
  SBP Day 21/4h postdose (metop. 25 mg) | 109.70 (NA) — NA=not calculated/1 subject | 115.50 (14.721) | 137.70 (NA) — NA=not calculated/1 subject
  SBP Day 21/8h postdose (metop. 25 mg): number analyzed (Participants) | 1 | 4 | 1
  SBP Day 21/8h postdose (metop. 25 mg) | 111.30 (NA) — NA=not calculated/1 subject | 118.43 (17.039) | 121.70 (NA) — NA=not calculated/1 subject
  SBP Day 21/12h postdose (metop. 25 mg): number analyzed (Participants) | 1 | 4 | 1
  SBP Day 21/12h postdose (metop. 25 mg) | 112.70 (NA) — NA=not calculated/1 subject | 122.00 (16.880) | 133.00 (NA) — NA=not calculated/1 subject
  SBP Day 15/predose (metop. 50 mg): number analyzed (Participants) | 3 | 3 | 2
  SBP Day 15/predose (metop. 50 mg) | 120.03 (14.048) | 123.47 (15.165) | 126.50 (16.263)
  SBP Day 15/2h postdose (metop. 50 mg): number analyzed (Participants) | 3 | 3 | 2
  SBP Day 15/2h postdose (metop. 50 mg) | 113.13 (8.501) | 117.47 (9.506) | 119.15 (18.173)
  SBP Day 15/4h postdose (metop. 50 mg): number analyzed (Participants) | 3 | 3 | 2
  SBP Day 15/4h postdose (metop. 50 mg) | 119.47 (18.742) | 121.67 (8.223) | 117.50 (19.092)
  SBP Day 15/8h postdose (metop. 50 mg): number analyzed (Participants) | 3 | 3 | 2
  SBP Day 15/8h postdose (metop. 50 mg) | 114.10 (20.301) | 121.00 (16.790) | 114.70 (5.657)
  SBP Day 15/12h postdose (metop. 50 mg): number analyzed (Participants) | 3 | 3 | 2
  SBP Day 15/12h postdose (metop. 50 mg) | 120.33 (15.216) | 122.23 (12.168) | 116.85 (9.687)
  SBP Day 18/predose (metop. 50 mg): number analyzed (Participants) | 3 | 6 | 1
  SBP Day 18/predose (metop. 50 mg) | 124.10 (15.650) | 115.55 (7.441) | 122.30 (NA) — NA=not calculated/1 subject
  SBP Day 18/2h postdose (metop. 50 mg): number analyzed (Participants) | 3 | 6 | 1
  SBP Day 18/2h postdose (metop. 50 mg) | 117.57 (9.416) | 108.90 (11.661) | 117.70 (NA) — NA=not calculated/1 subject
  SBP Day 18/4h postdose (metop. 50 mg): number analyzed (Participants) | 3 | 6 | 1
  SBP Day 18/4h postdose (metop. 50 mg) | 117.47 (6.486) | 113.12 (14.809) | 125.30 (NA) — NA=not calculated/1 subject
  SBP Day 18/8h postdose (metop. 50 mg): number analyzed (Participants) | 3 | 6 | 1
  SBP Day 18/8h postdose (metop. 50 mg) | 124.10 (13.028) | 123.28 (13.124) | 117.70 (NA) — NA=not calculated/1 subject
  SBP Day 18/12h postdose (metop. 50 mg): number analyzed (Participants) | 3 | 6 | 1
  SBP Day 18/12h postdose (metop. 50 mg) | 120.90 (12.819) | 110.22 (10.286) | 117.70 (NA) — NA=not calculated/1 subject
  SBP Day 21/predose (metop. 50 mg): number analyzed (Participants) | 3 | 4 | 3
  SBP Day 21/predose (metop. 50 mg) | 108.47 (4.895) | 111.10 (8.924) | 129.90 (14.626)
  SBP Day 21/2h postdose (metop. 50 mg): number analyzed (Participants) | 3 | 4 | 3
  SBP Day 21/2h postdose (metop. 50 mg) | 108.53 (5.654) | 107.15 (4.012) | 124.67 (8.793)
  SBP Day 21/4h postdose (metop. 50 mg): number analyzed (Participants) | 3 | 4 | 3
  SBP Day 21/4h postdose (metop. 50 mg) | 114.10 (4.004) | 108.18 (6.185) | 127.13 (12.044)
  SBP Day 21/8h postdose (metop. 50 mg): number analyzed (Participants) | 3 | 4 | 3
  SBP Day 21/8h postdose (metop. 50 mg) | 111.90 (1.929) | 108.28 (7.775) | 130.53 (15.747)
  SBP Day 21/12h postdose (metop. 50 mg): number analyzed (Participants) | 3 | 4 | 3
  SBP Day 21/12h postdose (metop. 50 mg) | 105.43 (1.401) | 112.08 (4.749) | 133.10 (14.674)
  SBP Day 15/predose (metop. 100 mg): number analyzed (Participants) | 3 | 6 | 3
  SBP Day 15/predose (metop. 100 mg) | 112.63 (6.429) | 114.93 (12.018) | 136.00 (22.203)
  SBP Day 15/2h postdose (metop. 100 mg): number analyzed (Participants) | 3 | 6 | 2
  SBP Day 15/2h postdose (metop. 100 mg) | 106.47 (7.679) | 107.40 (10.153) | 127.20 (21.920)
  SBP Day 15/4h postdose (metop. 100 mg): number analyzed (Participants) | 3 | 6 | 2
  SBP Day 15/4h postdose (metop. 100 mg) | 105.00 (6.000) | 111.70 (10.995) | 124.00 (15.556)
  SBP Day 15/8h postdose (metop. 100 mg): number analyzed (Participants) | 3 | 6 | 2
  SBP Day 15/8h postdose (metop. 100 mg) | 107.37 (4.619) | 113.60 (13.686) | 127.65 (12.233)
  SBP Day 15/12h postdose (metop. 100 mg): number analyzed (Participants) | 3 | 6 | 2
  SBP Day 15/12h postdose (metop. 100 mg) | 105.97 (3.215) | 107.37 (12.757) | 126.50 (13.011)
  SBP Day 18/predose (metop. 100 mg): number analyzed (Participants) | 1 | 2 | 3
  SBP Day 18/predose (metop. 100 mg) | 115.00 (NA) — NA=not calculated/1 subject | 125.35 (6.152) | 120.43 (5.353)
  SBP Day 18/2h postdose (metop. 100 mg): number analyzed (Participants) | 1 | 2 | 3
  SBP Day 18/2h postdose (metop. 100 mg) | 106.00 (NA) — NA=not calculated/1 subject | 121.50 (10.607) | 121.23 (0.681)
  SBP Day 18/4h postdose (metop. 100 mg): number analyzed (Participants) | 1 | 2 | 3
  SBP Day 18/4h postdose (metop. 100 mg) | 110.30 (NA) — NA=not calculated/1 subject | 122.85 (7.283) | 121.00 (1.480)
  SBP Day 18/8h postdose (metop. 100 mg): number analyzed (Participants) | 1 | 2 | 3
  SBP Day 18/8h postdose (metop. 100 mg) | 112.30 (NA) — NA=not calculated/1 subject | 116.20 (2.121) | 124.43 (5.518)
  SBP Day 18/12h postdose (metop. 100 mg): number analyzed (Participants) | 1 | 2 | 3
  SBP Day 18/12h postdose (metop. 100 mg) | 109.70 (99999) | 118.15 (6.859) | 118.90 (4.703)
  SBP Day 21/predose (metop. 100 mg): number analyzed (Participants) | 5 | 5 | 2
  SBP Day 21/predose (metop. 100 mg) | 123.12 (11.031) | 117.02 (3.710) | 115.30 (NA) — NA=not calculated/1 subject
  SBP Day 21/2h postdose (metop. 100 mg): number analyzed (Participants) | 5 | 5 | 1
  SBP Day 21/2h postdose (metop. 100 mg) | 118.42 (10.545) | 109.26 (8.021) | 110.00 (NA) — NA=not calculated/1 subject
  SBP Day 21/4h postdose (metop. 100 mg): number analyzed (Participants) | 5 | 5 | 1
  SBP Day 21/4h postdose (metop. 100 mg) | 122.94 (8.961) | 117.68 (7.477) | 112.70 (NA) — NA=not calculated/1 subject
  SBP Day 21/8h postdose (metop. 100 mg): number analyzed (Participants) | 5 | 5 | 1
  SBP Day 21/8h postdose (metop. 100 mg) | 124.00 (11.655) | 118.74 (12.817) | 117.00 (NA) — NA=not calculated/1 subject
  SBP Day 21/12h postdose (metop. 100 mg): number analyzed (Participants) | 5 | 5 | 1
  SBP Day 21/12h postdose (metop. 100 mg) | 123.60 (11.996) | 116.74 (10.827) | 117.70 (NA) — NA=not calculated/1 subject

12. Secondary Outcome: Trough Concentration (Ctrough) of Tesofensine on Day 13, Day 14, Day 15, Day 18, Day 21 and Day 23
Time Frame: Pre-dose on Day 13, Day 14 and Day 23. Pre-dose on Day 15, Day 18 and Day 21 is listed as Metoprolol 25 mg, Metoprolol 50 mg and Metoprolol 100 mg since metoprolol was administered in randomized order.
Population: Pharmacokinetic population required at least 1 quantifiable concentration, thus subjects discontinued before Day 13 were excluded. The number of participants listed below is the number of subjects with an assessment at the specified time point.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Cohort 1 (Tesofensine 0.25mg) | Cohort 2 (Tesofensine 0.50mg) | Cohort 3 (Tesofensine 0.75mg)
Number analyzed (Participants) | 9 | 14 | 7
ng/mL
  Day 13 | 3.293 (27.94) | 8.056 (35.33) | 12.20 (21.29)
  Day 14 | 3.471 (28.81) | 7.827 (35.67) | 12.10 (18.40)
  Day 23;: number analyzed (Participants) | 9 | 12 | 5
  Day 23; | 4.073 (30.23) | 8.569 (35.40) | 13.96 (28.60)
  Metoprolol 25 mg: number analyzed (Participants) | 9 | 13 | 6
  Metoprolol 25 mg | 3.377 (32.74) | 7.568 (30.37) | 11.96 (24.09)
  Metoprolol 50 mg: number analyzed (Participants) | 9 | 14 | 6
  Metoprolol 50 mg | 3.457 (27.58) | 7.940 (37.85) | 11.52 (23.62)
  Metoprolol 100 mg: number analyzed (Participants) | 9 | 13 | 6
  Metoprolol 100 mg | 3.322 (25.83) | 7.306 (29.61) | 12.21 (23.99)

13. Secondary Outcome: Maximum Serum Concentration (Cmax) of Metoprolol on Day 15, Day 18, and Day 21
Time Frame: Day 15, Day 18 and Day 21
Population: Pharmacokinetic (PK) population: All randomized subjects with at least 1 quantifiable tesofensine or metoprolol concentration and without major protocol deviations which could have influenced the PK.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg/L
Arm/Group | Cohort 1 (Tesofensine 0.25mg) | Cohort 2 (Tesofensine 0.50mg) | Cohort 3 (Tesofensine 0.75mg)
Number analyzed (Participants) | 9 | 13 | 6
μg/L
  Metoprolol 25 mg | 5.215 (93.04) | 6.402 (49.71) | 6.009 (45.95)
  Metoprolol 50 mg | 12.91 (61.51) | 14.91 (54.30) | 13.25 (32.13)
  Metoprolol 100 mg | 22.85 (55.83) | 25.83 (46.79) | 27.59 (51.38)

14. Secondary Outcome: Time to Cmax (Tmax) of Metoprolol on Day 15, Day 18, and Day 21
Time Frame: Day 15, Day 18 and Day 21
Population: as for outcome 13
Measure: Median (Full Range); unit: hours
Arm/Group | Cohort 1 (Tesofensine 0.25mg) | Cohort 2 (Tesofensine 0.50mg) | Cohort 3 (Tesofensine 0.75mg)
Number analyzed (Participants) | 9 | 13 | 6
hours
  Metoprolol 25 mg | 12.0 [8.0 to 12] | 8.03 [8.0 to 12] | 9.98 [8.0 to 12]
  Metoprolol 50 mg | 7.98 [4.0 to 12] | 8.02 [4.1 to 12] | 10.2 [8.0 to 12]
  Metoprolol 100 mg | 4.02 [4.0 to 23] | 8.00 [4.0 to 12] | 8.04 [8.0 to 12]

15. Secondary Outcome: Area Under the Concentration-time Curve From 0 to 24 h (AUC 0-24) of Metoprolol on Day 15, Day 18, and Day 21
Time Frame: Day 15, Day 18 and Day 21
Population: as for outcome 13
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*μg/L
Arm/Group | Cohort 1 (Tesofensine 0.25mg) | Cohort 2 (Tesofensine 0.50mg) | Cohort 3 (Tesofensine 0.75mg)
Number analyzed (Participants) | 9 | 13 | 6
h*μg/L
  Metoprolol 25 mg | 91.791 (87.70) | 105.41 (51.46) | 104.90 (54.76)
  Metoprolol 50 mg | 203.19 (65.50) | 240.92 (58.21) | 221.59 (28.47)
  Metoprolol 100 mg | 392.70 (67.88) | 458.35 (52.06) | 466.34 (45.85)

16. Secondary Outcome: Heart Rate (HR) Stratified by Metoprolol Concentration
Time Frame: Day before dosing (Days 14, 17, 20), dosing day (Days 15, 18, 21) and two days after dosing (Days 17, 20, 23)
Measure: Mean (Standard Deviation); unit: bpm
Arm/Group | Cohort 1 (Tesofensine 0.25mg) | Cohort 2 (Tesofensine 0.50mg) | Cohort 3 (Tesofensine 0.75mg)
Number analyzed (Participants) | 9 | 13 | 6
bpm
  Metoprolol 25 mg; Day before dosing | 73.8 (9.96) | 79.4 (8.13) | 82.2 (7.41)
  Metoprolol 25 mg; Dosing day | 71.1 (9.45) | 76.5 (7.68) | 80.0 (7.71)
  Metoprolol 25 mg; Two days after dosing | 76.8 (10.94) | 82.1 (8.88) | 85.7 (7.47)
  Metoprolol 50 mg; Day before dosing | 74.3 (9.62) | 78.7 (5.47) | 85.5 (7.92)
  Metoprolol 50 mg; Dosing day | 69.6 (9.40) | 73.9 (5.75) | 80.8 (7.83)
  Metoprolol 50 mg; Two days after dosing | 76.2 (10.06) | 82.1 (7.22) | 83.0 (7.11)
  Metoprolol 100 mg; Day before dosing | 75.2 (9.30) | 77.6 (5.47) | 81.2 (5.26)
  Metoprolol 100 mg; Dosing day | 69.2 (9.46) | 70.7 (6.05) | 73.6 (3.91)
  Metoprolol 100 mg; Two days after dosing | 76.6 (10.13) | 78.8 (4.26) | 84.4 (8.91)

17. Secondary Outcome: Change From Baseline Mean Heart Rate Over 24 Hours (M24HR) by Metoprolol Dose
Description: The difference in increase in M24HR caused by tesofensine alone (calculated as the difference between the M24HR at pre-tesofensine baseline and the mean of M24HR on Days 14, 17, 20 and 23) and the reduction in M24HR following each of the 3 metoprolol doses (M24HR on Day 15, 18 or 21).
Time Frame: From baseline to Day 23
Population: as for outcome 7
Measure: Mean (95% Confidence Interval); unit: bpm
Arm/Group | Cohort 1 (Tesofensine 0.25mg) | Cohort 2 (Tesofensine 0.50mg) | Cohort 3 (Tesofensine 0.75mg)
Number analyzed (Participants) | 9 | 13 | 6
bpm
  Metoprolol 25 mg: number analyzed (Participants) | 9 | 13 | 5
  Metoprolol 25 mg | -1.17 [-4.84 to 2.49] | 3.55 [0.34 to 6.77] | 6.97 [4.77 to 9.16]
  Metoprolol 50 mg | -2.99 [-6.63 to 0.65] | 0.88 [-2.34 to 4.11] | 7.98 [5.91 to 10.15]
  Metoprolol 100 mg: number analyzed (Participants) | 9 | 13 | 5
  Metoprolol 100 mg | -3.59 [-7.25 to 0.08] | -2.13 [-5.37 to 1.10] | 0.45 [-2.04 to 2.94]

18. Secondary Outcome: Mean of Triplicated QT Interval
Description: Mean of triplicated QT Interval
Time Frame: Day -1, Day 13 [pre-dose only], Day 14, Day 15, Day 17, Day 18, Day 20, Day 21 and Day 23
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: msec
Arm/Group | Cohort 1 (Tesofensine 0.25mg) | Cohort 2 (Tesofensine 0.50mg) | Cohort 3 (Tesofensine 0.75mg)
Number analyzed (Participants) | 9 | 16 | 12
msec
  Day -1/predose | 400.00 (23.654) | 398.08 (22.518) | 404.28 (31.567)
  Day -1/2h postdose | 381.83 (20.867) | 375.76 (15.028) | 386.66 (30.168)
  Day -1/4h postdose | 388.29 (27.746) | 385.91 (14.718) | 396.34 (28.389)
  Day -1/8h postdose | 395.78 (22.869) | 391.67 (16.588) | 395.12 (19.830)
  Day -1/12h postdose | 378.00 (26.099) | 385.30 (16.044) | 387.56 (28.855)
  Day 13/predose: number analyzed (Participants) | 9 | 14 | 7
  Day 13/predose | 404.14 (24.739) | 384.81 (13.394) | 390.59 (19.371)
  Day 14/predose: number analyzed (Participants) | 9 | 14 | 7
  Day 14/predose | 402.81 (28.425) | 396.81 (13.317) | 398.19 (16.649)
  Day 14/2h postdose: number analyzed (Participants) | 9 | 14 | 7
  Day 14/2h postdose | 392.37 (30.650) | 386.39 (18.472) | 383.24 (18.341)
  Day 14/4h postdose: number analyzed (Participants) | 9 | 14 | 7
  Day 14/4h postdose | 398.01 (30.117) | 385.48 (14.826) | 389.43 (18.661)
  Day 14/8h postdose: number analyzed (Participants) | 9 | 14 | 7
  Day 14/8h postdose | 396.82 (30.306) | 386.01 (16.595) | 389.64 (16.190)
  Day 14/12h postdose: number analyzed (Participants) | 9 | 14 | 7
  Day 14/12h postdose | 386.01 (28.991) | 379.14 (17.101) | 375.43 (19.292)
  Day 17/predose: number analyzed (Participants) | 9 | 13 | 7
  Day 17/predose | 405.10 (29.008) | 392.72 (19.161) | 393.53 (16.439)
  Day 17/2h postdose: number analyzed (Participants) | 9 | 13 | 6
  Day 17/2h postdose | 391.99 (31.469) | 377.69 (14.665) | 371.45 (14.113)
  Day 17/4h postdose: number analyzed (Participants) | 9 | 13 | 6
  Day 17/4h postdose | 400.02 (29.034) | 390.76 (16.704) | 382.88 (10.457)
  Day 17/8h postdose: number analyzed (Participants) | 9 | 13 | 6
  Day 17/8h postdose | 393.98 (25.616) | 384.11 (17.812) | 382.00 (9.674)
  Day 17/12h postdose: number analyzed (Participants) | 9 | 13 | 6
  Day 17/12h postdose | 378.51 (27.115) | 374.83 (10.381) | 368.33 (11.941)
  Day 20/predose: number analyzed (Participants) | 9 | 13 | 5
  Day 20/predose | 407.56 (28.115) | 390.52 (16.942) | 389.34 (16.182)
  Day 20/2h postdose: number analyzed (Participants) | 9 | 13 | 5
  Day 20/2h postdose | 390.23 (31.513) | 374.25 (13.470) | 376.68 (11.908)
  Day 20/4h postdose: number analyzed (Participants) | 9 | 13 | 5
  Day 20/4h postdose | 403.62 (31.402) | 384.93 (15.006) | 385.20 (22.302)
  Day 20/8h postdose: number analyzed (Participants) | 9 | 13 | 5
  Day 20/8h postdose | 398.67 (33.745) | 381.07 (13.220) | 392.26 (23.255)
  Day 20/12h postdose: number analyzed (Participants) | 9 | 13 | 5
  Day 20/12h postdose | 382.29 (35.547) | 368.41 (14.193) | 377.08 (17.626)
  Day 23/predose: number analyzed (Participants) | 9 | 12 | 5
  Day 23/predose | 403.10 (25.565) | 382.83 (19.770) | 387.76 (20.460)
  Day 23/2h postdose: number analyzed (Participants) | 9 | 12 | 5
  Day 23/2h postdose | 385.78 (24.461) | 371.06 (14.921) | 369.74 (18.183)
  Day 23/4h postdose: number analyzed (Participants) | 9 | 12 | 5
  Day 23/4h postdose | 394.16 (31.839) | 378.17 (19.816) | 386.14 (24.694)
  Day 23/8h postdose: number analyzed (Participants) | 9 | 12 | 5
  Day 23/8h postdose | 388.30 (28.021) | 375.13 (21.611) | 381.86 (19.204)
  Day 23/12h postdose: number analyzed (Participants) | 9 | 12 | 5
  Day 23/12h postdose | 376.07 (22.251) | 365.06 (19.474) | 371.62 (18.763)
  Day 15/predose (metop. 25 mg): number analyzed (Participants) | 3 | 4 | 3
  Day 15/predose (metop. 25 mg) | 403.10 (24.701) | 395.35 (5.735) | 384.00 (7.436)
  Day 15/2h postdose (metop. 25 mg): number analyzed (Participants) | 3 | 4 | 3
  Day 15/2h postdose (metop. 25 mg) | 376.23 (31.405) | 384.83 (7.265) | 374.67 (9.820)
  Day 15/4h postdose (metop. 25 mg): number analyzed (Participants) | 3 | 4 | 3
  Day 15/4h postdose (metop. 25 mg) | 392.20 (32.336) | 396.15 (9.293) | 384.23 (7.125)
  Day 15/8h postdose (metop. 25 mg): number analyzed (Participants) | 3 | 4 | 3
  Day 15/8h postdose (metop. 25 mg) | 399.33 (36.382) | 397.18 (15.108) | 388.67 (13.785)
  Day 15/12h postdose (metop. 25 mg): number analyzed (Participants) | 3 | 4 | 3
  Day 15/12h postdose (metop. 25 mg) | 396.43 (51.651) | 392.33 (12.747) | 378.20 (14.901)
  Day 18/predose (metop. 25 mg): number analyzed (Participants) | 5 | 5 | 2
  Day 18/predose (metop. 25 mg) | 405.48 (26.341) | 396.12 (15.396) | 363.35 (29.204)
  Day 18/2h postdose (metop. 25 mg): number analyzed (Participants) | 5 | 5 | 2
  Day 18/2h postdose (metop. 25 mg) | 394.94 (16.701) | 384.52 (10.925) | 381.35 (27.365)
  Day 18/4h postdose (metop. 25 mg): number analyzed (Participants) | 5 | 5 | 2
  Day 18/4h postdose (metop. 25 mg) | 412.14 (22.650) | 399.46 (17.580) | 386.00 (29.274)
  Day 18/8h postdose (metop. 25 mg): number analyzed (Participants) | 5 | 5 | 2
  Day 18/8h postdose (metop. 25 mg) | 411.86 (16.278) | 389.48 (15.161) | 378.30 (35.355)
  Day 18/12h postdose (metop. 25 mg): number analyzed (Participants) | 5 | 5 | 2
  Day 18/12h postdose (metop. 25 mg) | 401.06 (17.177) | 378.94 (16.214) | 364.65 (12.233)
  Day 21/predose (metop. 25 mg): number analyzed (Participants) | 1 | 4 | 1
  Day 21/predose (metop. 25 mg) | 368.70 (NA) — NA=not calculated/1subj. | 370.15 (13.164) | 384.00 (NA) — NA=not calculated/1subj.
  Day 21/2h postdose (metop. 25 mg): number analyzed (Participants) | 1 | 4 | 1
  Day 21/2h postdose (metop. 25 mg) | 376.70 (NA) — NA=not calculated/1subj. | 358.68 (12.613) | 375.30 (NA) — NA=not calculated/1subj.
  Day 21/4h postdose (metop. 25 mg): number analyzed (Participants) | 1 | 4 | 1
  Day 21/4h postdose (metop. 25 mg) | 358.70 (NA) — NA=not calculated/1subj. | 372.48 (8.330) | 376.70 (NA) — NA=not calculated/1subj.
  Day 21/8h postdose (metop. 25 mg): number analyzed (Participants) | 1 | 4 | 1
  Day 21/8h postdose (metop. 25 mg) | 386.00 (NA) — NA=not calculated/1subj. | 381.35 (18.034) | 395.30 (NA) — NA=not calculated/1subj.
  Day 21/12h postdose (metop. 25 mg): number analyzed (Participants) | 1 | 4 | 1
  Day 21/12h postdose (metop. 25 mg) | 372.70 (NA) — NA=not calculated/1subj. | 374.18 (12.217) | 366.00 (NA) — NA=not calculated/1subj.
  Day 15/predose (metop. 50 mg): number analyzed (Participants) | 3 | 3 | 2
  Day 15/predose (metop. 50 mg) | 408.20 (29.360) | 388.67 (17.402) | 372.30 (18.385)
  Day 15/2h postdose (metop. 50 mg): number analyzed (Participants) | 3 | 3 | 2
  Day 15/2h postdose (metop. 50 mg) | 386.67 (34.141) | 373.77 (15.187) | 380.35 (36.275)
  Day 15/4h postdose (metop. 50 mg): number analyzed (Participants) | 3 | 3 | 2
  Day 15/4h postdose (metop. 50 mg) | 396.87 (39.405) | 393.80 (12.387) | 375.00 (38.184)
  Day 15/8h postdose (metop. 50 mg): number analyzed (Participants) | 3 | 3 | 2
  Day 15/8h postdose (metop. 50 mg) | 405.57 (25.408) | 390.47 (3.281) | 393.00 (21.213)
  Day 15/12h postdose (metop. 50 mg): number analyzed (Participants) | 3 | 3 | 2
  Day 15/12h postdose (metop. 50 mg) | 392.63 (29.143) | 383.53 (0.404) | 378.00 (2.828)
  Day 18/predose (metop. 50 mg): number analyzed (Participants) | 3 | 6 | 1
  Day 18/predose (metop. 50 mg) | 396.20 (30.513) | 385.75 (18.862) | 381.30 (NA) — NA=not calculated/1subj.
  Day 18/2h postdose (metop. 50 mg): number analyzed (Participants) | 3 | 6 | 1
  Day 18/2h postdose (metop. 50 mg) | 387.13 (41.727) | 377.53 (7.314) | 346.70 (NA) — NA=not calculated/1subj.
  Day 18/4h postdose (metop. 50 mg): number analyzed (Participants) | 3 | 6 | 1
  Day 18/4h postdose (metop. 50 mg) | 410.03 (45.622) | 390.88 (16.413) | 358.00 (NA) — NA=not calculated/1subj.
  Day 18/8h postdose (metop. 50 mg): number analyzed (Participants) | 3 | 6 | 1
  Day 18/8h postdose (metop. 50 mg) | 406.20 (40.115) | 400.00 (27.450) | 396.00 (NA) — NA=not calculated/1subj.
  Day 18/12h postdose (metop. 50 mg): number analyzed (Participants) | 3 | 6 | 1
  Day 18/12h postdose (metop. 50 mg) | 399.77 (45.018) | 388.57 (19.421) | 374.70 (NA) — NA=not calculated/1subj.
  Day 21/predose (metop. 50 mg): number analyzed (Participants) | 3 | 4 | 3
  Day 21/predose (metop. 50 mg) | 406.43 (13.952) | 388.98 (15.647) | 378.43 (37.456)
  Day 21/2h postdose (metop. 50 mg): number analyzed (Participants) | 3 | 4 | 3
  Day 21/2h postdose (metop. 50 mg) | 391.57 (7.769) | 377.18 (22.436) | 371.57 (20.096)
  Day 21/4h postdose (metop. 50 mg): number analyzed (Participants) | 3 | 4 | 3
  Day 21/4h postdose (metop. 50 mg) | 402.87 (15.658) | 394.68 (21.586) | 388.90 (26.117)
  Day 21/8h postdose (metop. 50 mg): number analyzed (Participants) | 3 | 4 | 3
  Day 21/8h postdose (metop. 50 mg) | 419.30 (19.287) | 404.48 (14.866) | 388.23 (22.649)
  Day 21/12h postdose (metop. 50 mg): number analyzed (Participants) | 3 | 4 | 3
  Day 21/12h postdose (metop. 50 mg) | 407.80 (1.559) | 391.03 (18.953) | 379.10 (22.060)
  Day 15/predose (metop. 100 mg): number analyzed (Participants) | 3 | 6 | 2
  Day 15/predose (metop. 100 mg) | 381.10 (12.842) | 391.55 (16.914) | 397.65 (44.760)
  Day 15/2h postdose (metop. 100 mg): number analyzed (Participants) | 3 | 6 | 2
  Day 15/2h postdose (metop. 100 mg) | 387.10 (13.146) | 382.22 (10.369) | 388.65 (15.061)
  Day 15/4h postdose (metop. 100 mg): number analyzed (Participants) | 3 | 6 | 2
  Day 15/4h postdose (metop. 100 mg) | 419.77 (27,802) | 406.12 (17.056) | 406.65 (24.537)
  Day 15/8h postdose (metop. 100 mg): number analyzed (Participants) | 3 | 6 | 2
  Day 15/8h postdose (metop. 100 mg) | 419.33 (10.081) | 400.45 (27.301) | 414.65 (10.394)
  Day 15/12h postdose (metop. 100 mg): number analyzed (Participants) | 3 | 6 | 2
  Day 15/12h postdose (metop. 100 mg) | 414.43 (5.954) | 396.68 (14.125) | 398.00 (18.809)
  Day 18/predose (metop. 100 mg): number analyzed (Participants) | 1 | 2 | 3
  Day 18/predose (metop. 100 mg) | 389.30 (NA) — NA=not calculated/1subj. | 391.00 (15.556) | 380.90 (16.536)
  Day 18/2h postdose (metop. 100 mg): number analyzed (Participants) | 1 | 2 | 3
  Day 18/2h postdose (metop. 100 mg) | 371.30 (NA) — NA=not calculated/1subj. | 375.00 (14.566) | 374.00 (14.117)
  Day 18/4h postdose (metop. 100 mg): number analyzed (Participants) | 1 | 2 | 3
  Day 18/4h postdose (metop. 100 mg) | 380.70 (NA) — NA=not calculated/1subj. | 392.65 (20.718) | 391.53 (16.762)
  Day 18/8h postdose (metop. 100 mg): number analyzed (Participants) | 1 | 2 | 3
  Day 18/8h postdose (metop. 100 mg) | 386.00 (NA) — NA=not calculated/1subj. | 405.00 (21.213) | 392.87 (18.329)
  Day 18/12h postdose (metop. 100 mg): number analyzed (Participants) | 1 | 2 | 3
  Day 18/12h postdose (metop. 100 mg) | 369.30 (NA) — NA=not calculated/1subj. | 393.00 (7.071) | 382.87 (20.429)
  Day 21/predose (metop. 100 mg): number analyzed (Participants) | 1 | 2 | 3
  Day 21/predose (metop. 100 mg) | 406.80 (39.537) | 387.20 (14.916) | 390.70 (NA) — NA=not calculated/1subj.
  Day 21/2h postdose (metop. 100 mg): number analyzed (Participants) | 5 | 5 | 1
  Day 21/2h postdose (metop. 100 mg) | 383.60 (37.938) | 374.78 (16.698) | 410.70 (NA) — NA=not calculated/1subj.
  Day 21/4h postdose (metop. 100 mg): number analyzed (Participants) | 5 | 5 | 1
  Day 21/4h postdose (metop. 100 mg) | 400.78 (38.353) | 396.24 (17.208) | 428.70 (NA) — NA=not calculated/1subj.
  Day 21/8h postdose (metop. 100 mg): number analyzed (Participants) | 5 | 5 | 1
  Day 21/8h postdose (metop. 100 mg) | 410.94 (38.128) | 399.74 (24.355) | 428.70 (NA) — NA=not calculated/1subj.
  Day 21/12h postdose (metop. 100 mg): number analyzed (Participants) | 5 | 5 | 1
  Day 21/12h postdose (metop. 100 mg) | 393.48 (38.721) | 387.60 (16.030) | 402.00 (NA) — NA=not calculated/1subj.

19. Secondary Outcome: Use of Concomitant Medication From 30 Days Prior to Screening Until Day 50
Description: Any medicinal product, prescribed or over-the-counter (OTC), including herbal and other non-traditional remedies, was considered a concomitant medication.
Time Frame: 30 days prior to Screening until the Safety Follow-up phone call, up to Day 50
Measure: Number; unit: Count of participants
Arm/Group | Cohort 1 (Tesofensine 0.25mg) | Cohort 2 (Tesofensine 0.50mg) | Cohort 3 (Tesofensine 0.75mg)
Number analyzed (Participants) | 9 | 16 | 12
Count of participants
  ACETYLSALICYLIC ACID/concomitant | 1 | 1 | 0
  BEPANTHEN/concomitant | 2 | 0 | 0
  PARACETAMOL/concomitant | 1 | 2 | 1
  ANAESTHETICS, LOCAL/concomitant | 0 | 1 | 0
  IBUPROFEN/concomitant | 0 | 2 | 1
  METOPROLOL TARTRATE/concomitant | 0 | 1 | 0
  PANTOPRAZOLE/concomitant | 0 | 1 | 0
  UNACID [AMPICILLIN SODIUM;SULBACTAM SODIUM]/conco. | 0 | 1 | 0
  IBUPROFEN/prior | 0 | 1 | 0
  FOLIC ACID/concomitant | 0 | 1 | 0
  METEX [METHOTREXATE SODIUM]/concomitant | 0 | 1 | 0
  PREDNISOLONE/concomitant | 0 | 1 | 0
  METOPROLOL SUCCINATE/concomitant | 0 | 1 | 0
  HALOPERIDOL/concomitant | 0 | 0 | 1
  LORAZEPAM/concomitant | 0 | 0 | 1
  METOCLOPRAMIDE/concomitant | 0 | 0 | 1
  RISPERIDON BETA/concomitant | 0 | 0 | 1
  PARACETAMOL/prior | 0 | 0 | 1

ADVERSE EVENTS:
Time Frame: From first dose of study drug through Day 50
Description: Adverse events are reported per tesofensine dose group. Differentiation per metoprolol dose could not be delineated.
Arm/Group | Cohort 1 (Tesofensine 0.25mg) | Cohort 2 (Tesofensine 0.50mg) | Cohort 3 (Tesofensine 0.75mg)
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/16 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/9 | 1/16 | 1/12
Other Adverse Events (participants affected / at risk) | 7/9 | 15/16 | 12/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 (Tesofensine 0.25mg) (N=9) | Cohort 2 (Tesofensine 0.50mg) (N=16) | Cohort 3 (Tesofensine 0.75mg) (N=12)
Hypomania (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1)
Nervous system disorder (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Impulse-control disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 (Tesofensine 0.25mg) (N=9) | Cohort 2 (Tesofensine 0.50mg) (N=16) | Cohort 3 (Tesofensine 0.75mg) (N=12)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Atrial tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1)
Palpitations (Cardiac disorders) | 4 (7) | 7 (8) | 5 (8)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 2 (2) | 1 (1)
Ventricular extrasystoles (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Foreign body sensation in eyes (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Vision blurred (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Visual impairment (Eye disorders) | 1 (1) | 1 (2) | 2 (2)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1) | 2 (2) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 5 (5) | 2 (2)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Lip swelling (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 5 (5) | 1 (1)
Asthenia (General disorders) | 0 (0) | 1 (1) | 1 (1)
Chest discomfort (General disorders) | 1 (1) | 2 (2) | 0 (0)
Energy increased (General disorders) | 0 (0) | 1 (1) | 0 (0)
Exercise tolerance (General disorders) | 0 (0) | 2 (2) | 0 (0)
Fatigue (General disorders) | 0 (0) | 2 (2) | 1 (1)
Feeling abnormal (General disorders) | 0 (0) | 0 (0) | 3 (4)
Feeling cold (General disorders) | 0 (0) | 1 (1) | 0 (0)
Feeling hot (General disorders) | 0 (0) | 1 (1) | 0 (0)
Feeling of relaxation (General disorders) | 0 (0) | 1 (1) | 0 (0)
Mucosal dryness (General disorders) | 0 (0) | 2 (2) | 0 (0)
Thirst (General disorders) | 0 (0) | 1 (1) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Blood pressure increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Blood pressure systolic increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 3 (3) | 11 (11) | 9 (9)
Muscle rigidity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Muscle tightness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Aphasia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Coordination abnormal (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Disturbance in attention (Nervous system disorders) | 1 (1) | 3 (3) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 3 (5) | 3 (4)
Dizziness exertional (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Dizziness postural (Nervous system disorders) | 2 (2) | 1 (1) | 2 (2)
Dysarthria (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0)
Dyskinesia (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Facial neuralgia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Head discomfort (Nervous system disorders) | 0 (0) | 0 (0) | 1 (2)
Headache (Nervous system disorders) | 4 (7) | 5 (5) | 6 (6)
Parosmia (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Psychomotor hyperactivity (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Psychomotor skills impaired (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Sensory disturbance (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 3 (3) | 3 (3)
Tension headache (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Tremor (Nervous system disorders) | 1 (1) | 3 (4) | 1 (1)
Abnormal dreams (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Agitation (Psychiatric disorders) | 1 (1) | 2 (2) | 2 (2)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Confusional state (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Euphoric mood (Psychiatric disorders) | 1 (1) | 6 (6) | 4 (4)
Fear (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Hallucination (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1)
Hypomania (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Illusion (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 3 (3) | 3 (3)
Irritability (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1)
Listless (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Mood altered (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Mood swings (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Restlessness (Psychiatric disorders) | 1 (1) | 1 (1) | 0 (0)
Sleep disorder (Psychiatric disorders) | 0 (0) | 7 (7) | 5 (6)
Tension (Psychiatric disorders) | 2 (2) | 4 (4) | 2 (2)
Thinking abnormal (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Tic (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Pollakisuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Breast discomfort (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Breast tenderness (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Menstrual discomfort (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pharyngeal disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Yawning (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 1 (1)
Hot flush (Vascular disorders) | 0 (0) | 1 (2) | 2 (2)
Rash (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Catheter site pain (General disorders) | 1 (1) | 0 (0) | 0 (0)
Chest pain (General disorders) | 1 (2) | 1 (1) | 0 (0)
Medical device site reaction (General disorders) | 3 (3) | 0 (0) | 0 (0)
Arthropod bite (Injury, poisoning and procedural complications) | 2 (2) | 1 (1) | 0 (0)
Epicondylitis (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Trigger finger (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Dysaesthesia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Taste disorder (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Finger repair operation (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2018-06-14): https://cdn.clinicaltrials.gov/large-docs/19/NCT03488719/Prot_000.pdf
  • Statistical Analysis Plan (2019-07-05): https://cdn.clinicaltrials.gov/large-docs/19/NCT03488719/SAP_001.pdf